## Official Title Neuromodulation of Cognition in Older Adults

NCT number NCT02137122

Document Date 5/13/2019

#### Protocol # 201400328

## 1. Project Title

Neuromodulation of Cognition in Older Adults: The Stimulated Brain Study

## 2. Investigator(s):

Adam J. Woods, PhD Ron Cohen, PhD Michael Marsiske, PhD Samuel Wu, PhD Steve Anton, PhD Eric Porges, PhD Marco Pahor, MD Song Lai, PhD

Andrew O'Shea M.Sc.: Study Coordinator

Nicole Nissim, M.S.

Keyanni Joy Johnson

Roxanne Rezaei, B.A.

Jessica Kraft, M.A.

Aprinda Indahlastari, Ph.D

Cindy Hernandez, B.S.

Alexa Chen, B.A.

Kathleen Frost, B.S.

Kelsey Traeger, B.S.

Kristin Calfee, B.A.

Alexander Albizu, B.S.

Steven DeKosky, M.D.

Emanuel Boutzoukas, B.S.

Daniela Carballo

Nicole Evangelista

Hanna Hausman, B.A.

Sam Vrinios

Margaret Meldrum

Sean Perryman, B.A.

Vanessa Dominguez, B.S.

Matt Fillingim

#### 3. Abstract:

The current study will investigate methods for enhancing cognitive training (CT) effects in healthy older adults by employing a combination of interventions facilitating neural

Protocol IRB #201400328 IRB version 03.09.04 PI version 5/13/2019

plasticity and optimizing readiness for learning. Adults over the age of 65 represent the fastest growing group in the US population. As such, age-related cognitive decline represents a major concern for public health. Recent research suggests that cognitive training in older adults can improve cognitive performance, with effects lasting up to 10 years. However, these effects are typically limited to the tasks trained, with little transfer to other cognitive abilities or everyday skills. A pilot randomized clinical trial will examine the individual and combined impact of pairing cognitive training with transcranial direct current stimulation (tDCS). tDCS is a method of non-invasive brain stimulation that directly stimulates brain regions involved in active cognitive function and enhances neural plasticity when paired with a training task. We will compare changes in cognitive and brain function resulting from CT combined with active tDCS versus CT combined with sham tDCS using a comprehensive neurocognitive, clinical, and multimodal neuroimaging assessment of brain structure, function, and metabolic state. Functional magnetic resonance imaging (FMRI) will be used to assess brain response during working memory, attention, and memory encoding; the active cognitive abilities trained by CT. Proton magnetic resonance spectroscopy (MRS) will assess cerebral metabolites, including GABA concentrations sensitive to neural plasticity.

## We hypothesize that:

- 1) tDCS will enhance neurocognitive function, brain function, and functional outcomes from CT, with combined CT and tDCS providing the most benefit;
- 2) Effects of tDCS on CT will be maintained up to 3 months following training
- 3) Neuroimaging biomarkers of cerebral metabolism, neural plasticity (GABA concentrations) and functional brain response (FMRI) during resting vs. active cognitive tasks will predict individual response to tDCS.

To date, no studies have examined combined intervention strategies using CT or optimization of learning and functional status through facilitation of active versus resting brain states in the elderly. The present study will provide a unique window into critical mechanisms for combating cognitive decline in a rapidly aging US population and novel methods for counteracting this looming public health crisis.

## 4. Background:

**4.1. Public Health / Clinical Significance**: **1)** Increased life expectancy has resulted in a marked increase of the older population. **2)** Cognitive changes occur with advanced age that affect functional and health status. **3)** While Alzheimer's and related neurodegenerative diseases cause the most dramatic cognitive disturbances in the elderly, cognitive aging occurs even among people considered to be neurologically healthy. **4)** Even mild neurocognitive disturbances affect people's daily functioning, health status, and quality of life. **5)** Alterations of brain structure and function occur as people reach advanced age, along with cerebral metabolic changes, that are associated with neurocognitive decline. **6)** Our preliminary data suggests that baseline cerebral metabolite (MRS) and functional neuroimaging (FMRI) indices are associated with baseline neurocognitive functioning and predictive of subsequent age-related cognitive decline and brain disturbances. **7)** There is a paucity of preventive and treatment

interventions for averting cognitive aging and enhancing cognitive function. **8)** Certain cognitive training (CT) approaches improve specific areas of cognitive performance, although their relative efficacy and mechanisms of action are not well understood. **9)** Most CT approaches do not generalize well to cognitive abilities beyond those being trained or to everyday functional abilities. Efforts are needed to improve the generalizability of CT. **10)** Methods exist which could potentiate CT (e.g., tDCS), but they have not been rigorously tested in RCTs.

**4.2. Scientific significance. 1)** While there is evidence that CT can improve cognitive functioning, the underlying mechanisms are not well understood. 2) The efficacy of CT likely is dependent on the plasticity of neural systems. 3) Evidence that certain types of neurochemical, electrical and behavioral stimulation potentiates synaptic plasticity and enhances learning has been demonstrated in laboratory animals. It is important to be able to measure these changes in humans during the course of learning such as that occurring with CT. Yet, in vivo human studies of these effects are difficult for obvious reasons. 4) Functional (FMRI) and cerebral metabolic (MRS) neuroimaging indirectly assess changes in neural plasticity during cognitive tasks. Recent developments in MRS enable Gama Amino butyric Acid (GABA), the primary inhibitory neurotransmitter and an essential neurotransmitter for synaptic communication and associative formation, to be measured from brain regions of interest (ROIs) 12. GABA concentrations predict attentional control 1 and sensory discrimination 3,4, decrease with age<sup>5</sup> and yet demonstrate long-term increase with learning interventions. <sup>2,6</sup>. Functional connectivity measured by FMRI provides another potentially powerful approach for measuring these changes. Yet, these neuroimaging approaches have been employed to only a very limited extent in studies of the mechanisms of CT. Studies employing neuroimaging to assess CT outcome are needed. 5) Many open questions exist regarding the brain's structural and functional connectivity in relationship to regional cerebral metabolites. Achieving better understanding of these relationships is important, since cerebral metabolic alterations may contribute neuropathology and perhaps even normal cognitive aging. 6) Extensive research exists for each of these neuroimaging modalities in isolation for various diseases, but multimodal studies employing these approaches simultaneously are less common, particularly in studies of normal aging or CT. 7) Various CT approaches exist, but only a few have been tested and shown to be effective in larger scale clinical trials (e.g., UFOV, dual N-back training). RCTs are needed to test the relative efficacy of these CT approaches, and whether there is value in using them in combination. 8) Brain stimulation may potentiate neural plasticity based on animal studies. Most of these approaches have yet to be tested in conjunction with CT in humans. 9) It is unclear whether optimal CT benefit is achieved by bolstering activation of brain regions necessary for the tasks to be performed. 10) Individual differences exist in the ability of people to benefit from CT. These differences are not well understood. We will examine neuroimaging and behavioral factors that predict CT outcome and that may account for these individual differences. 11) State-of-the-art neuroimaging analysis methods may yield insights into interactions among brain networks/systems, and ways to optimally integrate structural and functional connectivity with cerebral MRS and cognitive outcomes. 12) We will employ state-of-the-art

statistical methods, extending predictive modeling and causal inference approaches for neuroimaging.

## 4.3. Clinical and scientific background.

- **4.3.1.** Cognitive aging and dysfunction affects health status, Quality of Life (QOL), and functional capacity. Brain dysfunction resulting from neurodegenerative disease or other medical condition adversely affects overall health status.<sup>7-11</sup> Even mild cognitive deficits affect QOL, diet, physical activity and other health behaviors, <sup>10,12,13</sup> and are often stronger predictors of health outcomes than other physical factors, <sup>7</sup> but typically receive less clinical attention. Accordingly, cognitive aging has considerable functional relevance.
- **4.3.2. Cognitive training.** Various CT approaches enhance cognitive functioning in the elderly and remediate cognitive disorders. While improvements in cognitive performance are reported in many studies, this research suffers from a lack of wellconducted RCTs designed to determine the specific factors contributing to cognitive improvements. However, several approaches are effective in improving cognitive performance in the context of large RCTs. The ACTIVE study showed that CT improved cognitive performance and resulted in some generalization to other functional abilities. **4.3.3. Benefits of cognitive training.** Various CT approaches exist. While improved cognitive performance is often reported, this research has suffered from a lack of wellcontrolled RCTs, experimental designs that did not enable the basis for effects to be determined, and limited transfer of training. 14-18 Yet, findings over the past decade (e.g., ACTIVE) suggest that certain CT approaches are effective for enhancing cognitive aging. 17,19-36 Significant cognitive and functional improvements occur in laboratory and home-based CT studies. 19,23,31,37-41 Effect sizes generally exceed d=1.0 immediately after CT, and even after 10 years ( $\eta^2 > 0.6$ .). In ACTIVE,  $^{22,24,32,36,42}$  people receiving CT outperformed those who were untrained, with normal cognitive aging attenuated. We considered and selected CT approaches based on consensus of our study team (Woods, Marsiske, Edwards, Czaja, et al.), and evidence supporting their effectiveness. Three types of CT training have been particularly effective in studies by our group and others: 1) UFOV; 2) N-back Working Memory; 3) Attention-arousal training, all available in the PositScience BrainHQ suite (See Miscellaneous Attachments for detailed descriptions/samples of each game.)

## Attention/Speed of Processing

- 1. Hawk Eye- works on visual precision, which helps the brain perceive what you see quickly and accurately so that you can recall it better.
- Divided Attention- requires the brain to focus in on and react to particular details—matching colors, shapes, and/or fill patterns—while at the same time dismissing competing information.
- 3. Target Tracker- is designed to help build divided attention by requiring you to track several items moving around your screen at the same time
- 4. Double Decision\_requires visual search and selective attention to peripheral objects among distractors. Difficulty gradually increases relative to object similarity, presentation rate, and distractor complexity and eccentricity.

## Working Memory

- To Do List Training- the brain hears a set of instructions, then uses its memory of those instructions to follow them in order. The instructions get longer and more complex over time at the task, making greater demands of your working memory systems.
- 2. Memory Grid Auditory processing is one of the most important building blocks of memory. Only when you take in information with crystal clarity can the brain store it accurately and recall it clearly later. In Memory Grid, the task is to match cards representing syllables together.
- 3. Auditory Aces- Participant will be presented with auditory information about playing cards. The information is presented one card at a time. The task is to decide if the current card information matches the card information presented a specific number of steps back in the sequence.
- 4. Card Shark- N-back working memory task that varies on whether the current target matches stimuli presented 0-n steps before and presentation speed, leading to increased difficulty, 44,45 and age-sensitivity 46.
- **4.3.4. Generalization and functional outcome.** Training transfer has been most studied and shown on UFOV. In ACTIVE, ten-year maintenance of UFOV training effects occurred with evidence of substantial transfer at 5 and 10 years. UFOV training resulted in fewer self-reported limitations of everyday activities, 24 higher locus of control <sup>30</sup> and perceived health-related quality of life, <sup>68</sup> better subjective health, <sup>29</sup> and less depression.<sup>27</sup> <sup>68</sup> At ten years, UFOV-trained people still reported less limitation in daily activities<sup>36</sup>. Self-reported driving cessation and archival accident records indicated lower odds of crashes and driving cessation for UFOV-trained elders at three, 25 five, 28 and ten-years post training.35 In other RCTs involving greater sustained adaptive CT dosages (similar to the currently proposed study) superior performance and reaction times were found on a driving-simulator and also for instrumental activities of daily living (look up phone numbers, read pill bottles, etc.).<sup>23</sup> For the other two intervention components, near transfer to other cognitive tasks has been shown. N-back training transfers to matrix reasoning<sup>44</sup> and to sustained attention and self-reported cognitive function in older adults for at least three months post training. 48 Tonic/phasic attention training transfers to spatial selective attention and the temporal distribution of attention (attentional blink).66
- **4.3.5. Brain stimulation to potentiate training.** Since the pioneering work of Penfield, it has been recognized that sensory, motor and cognitive functions could be altered via electrical stimulation of specific brain regions. In laboratory animals, brain stimulation represented an alternative approach to experimental lesions, enabling both the potentiation and inhibition of neural activity depending on where in the brain stimulation was applied. Until recently, most human brain stimulation studies involved neurosurgically implanted electrodes, which has obvious limitations for general clinical use. **Transcranial direct current stimulation (tDCS)** is a non-invasive brain

stimulation method that alters the sub threshold membrane potential of neurons. facilitates neural plasticity and learning, and increases regional blood flow while modulating local GABA concentrations during stimulation. <sup>69-89</sup> During tDCS, a weak electrical current is applied to the scalp that penetrates skin, bone, CSF and the meninges to stimulate underlying cortical and subcortical tissue. 90-95 tDCS applied to dysfunctional cortical regions improves performance on a variety of cognitive tasks. 96-99 Bilateral tDCS to the frontal cortices improves decision-making, attention and working memory performance in older adults. 100-103 Improvements from a single session of tDCS have been shown to last for up to five years in healthy adults. 104-108 Small pilot RCTs (n=20/group) pairing CT with bilateral frontal tDCS show significant and lasting improvement in older adults experiencing declining cognitive function. 108-112 Maintenance of these tDCS and CT effects have been shown to last beyond one year. 104,105,107,108,110 These studies demonstrate that CT combined with tDCS leads to lasting improvement in CT effectiveness for older adults and patients. Research suggests that increased regional blood flow and decreased GABA concentrations during tDCS facilitate the brain's neural plastic response to paired training tasks. 75,80,83,84,89,113-117 Pairing CT with tDCS to combat age-related cognitive decline holds great promise for older adults.

- **4.3.6. Age-associated brain changes.** It is well known that with advanced age, humans are vulnerable to neurodegenerative diseases that cause brain pathology, usually evident on post-mortem autopsy. Though less pervasive, neuropathology is also relatively common in elderly adults without documented brain disease. A.3.6.1. **Age-associated brain change on structural neuroimaging.** Changes in structural brain volume and morphometry on MRI, along with specific abnormalities, occur with advanced age, particularly when there is vascular co-morbidity. Raz et al. showed cortical and subcortical volume loss of .5 -4% per year across different cortical and subcortical regions in older adults without overt brain disease. Respectively when the per year across the lifespan in past large international studies.
- **4.3.6.3. Functional neuroimaging** provides a potentially powerful method for assessing healthy and abnormal brain functioning (see Cohen and Sweet, for a review<sup>168</sup>). FMRI is noninvasive, can be used in conjunction with structural MRI and MRS, and is sensitive to functional brain abnormalities. 153,157,169-179 It holds promise as a biomarker of cognitive aging, neural plasticity, and cognitive improvements following CT. Age-associated alterations in brain activation on FMRI during both rest state and active cognitive tasks have been demonstrated in many past studies. Unfortunately, the clinical potential of FMRI has yet to be fully realized, in part because many different paradigms have been employed across studies. Furthermore, longitudinal change in BOLD response as a function of aging has been examined in relatively few studies, and almost no large RCTs. Reduced cognitive reserve with aging has been linked to a number of FMRI effects, including HAROLD and PASA. 180-183 Chang et al. showed that cognitive reserve influences FMRI activation, with a reduced "dynamic range" of BOLD response during tasks relative to rest explaining this effect. 184-190 The concept of dynamic range is both important and useful, and will be discussed in greater detail when reviewing preliminary data (C4). ERP measures the speed at which the brain processes

cognitive information. These measures will provide markers of improvement in the temporal processing of information, a key element altered with age.

4.3.6.4. Cerebral metabolites (MRS): Proton MRS, which is sensitive to chemical compounds containing hydrogen, useful for measuring brain metabolites, including N-Acetyl Aspartate (NAA), choline (Cho), myo-inositol (MI), creatine (Cr), and glutamateglutamine complex (Glx). Our group and others have shown that MRS abnormalities occur among people with a variety of age-related brain disorders, including neurodegenerative disease, cerebrovascular disease, and HIV<sup>191-206</sup>, with reduced NAA and elevated MI associated with cognitive dysfunction and conversion to dementia. Elevated Cho and MI reflect inflammatory processes and glial and cell membrane disturbances, and are differentially associated with cognitive performance, clinical status, and also cortical, subcortical, and white matter volumes on MRI<sup>204-211</sup>. Thus, MRS is predictive of clinically significant neurocognitive dysfunction. 206,208-210 GABA, the brain's principle inhibitory neurotransmitter, <sup>212</sup> is essential for synaptic communication and regulation of neuronal excitability, <sup>213</sup> and neural plasticity. <sup>214-218</sup> It plays a key role in learning and memory<sup>219-235</sup> and modulates other behavioral and affective functions, including executive control and attention. <sup>236-238</sup> Decreased cerebral GABA occurs with advanced age, <sup>219,223,227,230</sup> and GABA dysregulation occurs in neurological and psychiatric conditions. 49,239-267 GABA delivered to the frontal cortex and hippocampus in animals facilitates cognitive and working memory performance. GABA can now be reliability measured using proton MRS, 5,268-273 based on seminal work by Edden (consultant). 274-278 GABA provides an in vivo biomarker of neural plasticity in brain ROIs important for the cognitive functions to be trained in our study. 276 84



A.3.8. Summary and Conceptual Model. Age-associated functional, structural and metabolic brain changes occur, even in the absence of frank neurodegenerative disease. CT holds promise for reducing the adverse effects of cognitive aging, enhancing neural plasticity, cognitive efficiency, functional capacity, and quality of life. In theory, CT benefits could be augmented by coupling it with other interventions that either

increase neural plasticity. Yet, relatively few of these approaches have been tested in RCTs, and the mechanisms underlying their effects are largely unknown. Even less is known about the combined effects of CT with tDCS. Our preliminary data provides strong support for CT to combat cognitive aging, and also for the effects of tDCS on cognition and brain function. We hypothesize that CT leads to improvements in neural plasticity (GABA MRS) and functional brain response (FMRI). In turn, this can lead to improved cerebral metabolic health and structural brain preservation. Coupling CT with tDCS will increase neural plasticity in brain areas important for working memory, focused attention, and executive control, improve effectiveness of CT, and ultimately cognitive health (see Figure 1 for conceptual model).

## 5. Specific Aims:

Age-related cognitive decline has become a major public health concern. As the population ages, the number of older adults experiencing cognitive and functional disturbances has increased. There is currently a paucity of effective interventions to prevent or treat cognitive decline or to enhance brain function in the elderly. The proposed study will recruit a cohort from the state with the highest growth of older adults. We will employ an adaptive randomized clinical trial (RCT) to test whether the benefits of cognitive training (CT) can be enhanced by a combined adjunctive intervention aimed at increasing neural plasticity and optimizing readiness for learning: transcranial direct current stimulation (tDCS).

Current CT approaches have been shown to improve performance on trained tasks, with effects lasting up to ten years 32,33,36,279,280. However, generalization of effects to other cognitive domains and everyday functioning has been a problem in the past. There is now compelling evidence that the elderly do experience functional improvements that persist long after initial training, though peoples' ability to derive such benefits varies. Combined interventions have rarely been examined and methods aimed at increasing neural plasticity and optimizing readiness for learning are only now beginning to be explored. The proposed study will test one theoretical approach for facilitating and optimizing CT effects on functional outcome. We will use an adjunctive physiological method to further stimulate task-related brain regions, directly enhancing neural responsivity/plasticity and ultimately learning. While theoretical rationales exist for each of these approaches, no studies to date have shown whether adjunctive administration can optimize learning and functional status in the elderly.

A randomized clinical trial will enroll 90 participants. Cognitively healthy elderly adults, age 65-90 will undergo either a CT intervention in combination with transcranial direct current brain stimulation (tDCS) or sham tDCS control. The CT intervention will employ a suite of adaptive training tasks from the POSIT Science Brain HQ<sup>281</sup>; a well validated CT method for enhancing cognitive functioning in the elderly. Participants will receive tDCS or sham/placebo prefrontal stimulation administered during training.

Participants will be assessed at baseline, after CT (2 weeks), and at 3-month follow-up. At each time point, a comprehensive neurocognitive, clinical and multimodal neuroimaging assessment of brain function, metabolic state, and brain structure will be conducted.

FMRI will be used to assess brain response during working memory, attention and memory encoding. Proton magnetic resonance spectroscopy (MRS) will assess cerebral metabolites, including gamma-aminobutyric acid (GABA) concentrations, sensitive to neural plasticity in task-associated brain regions.

The central hypothesis of this proposal is that tDCS will increase neural plasticity in task associated brain regions, facilitating effectiveness of CT and transfer to everyday function.

- **Aim 1.** Determine whether neurocognitive improvement and longer-term functional outcome (as measured by "ecological assessment") are better when CT is coupled with tDCS, an intervention that will increase neural plasticity and augment training effects.
  - **H1.1.** Active tDCS combined with CT will amplify effects of CT on measures of attention, working memory, executive functioning, and learning efficiency, while sham tDCS will not.
  - **H1.2.** Active tDCS will enhance near and far transfer of CT, but sham will not evidence near or far transfer.
- **Aim 2.** Determine whether CT combined with tDCS leads to greater functional and metabolic brain changes (FMRI, MRS). Effects will parallel Aim 1.
  - **H2.1.** Combined CT + tDCS will potentiate decrease activation in working memory and attentional (dorsolateral prefrontal cortex, medial frontal cortex, inferior parietal lobe, supplementary motor association cortex) brain systems, reflecting increased neural efficiency, while CT + sham tDCS will not. **H2.2** Cerebral metabolite alterations will occur secondary to CT and tDCS, with long-term increase in GABA and *N*-acetyl aspartate (NAA) concentrations, and decreased choline (Cho) and myoinositol (MI) concentrations in the frontal cortex and posterior parietal cortex. CT and tDCS will modulate MRS GABA in frontal areas. These effects will be specific to CT.

**Secondary aim.** We will examine which baseline factors (e.g., clinical, demographic, neuroimaging, cognitive) best predict individual differences in outcome.

#### 6. Research Plan:

- **6.1. Experimental design.** This study employs a randomized trial design with 90 participants. One factor with two levels [Factor 1 = stimulation type (active or sham) yields two cells. Thus, participants will be assigned to one of two conditions:
- 1: Active tDCS + CT
- 2: Sham tDCS + CT

CT has previously been established with strong effects on cognitive and functional outcomes. Some small clinical trials showed small to medium effects of tDCS in conjunction with CT.

Participants will be assessed at three primary time points during the study, plus one screening visit on the front end to be sure they meet all inclusion criteria for the study:

- 1) Informed Consent and Screening Visit
- 2) Assessment Visit #1- baseline pre-training;
- 3) Assessment Visit #2- post-2 weeks
- 4) Assessment Visit #3- three month follow-up after all training (see Figure below for summary).

This design will enable longitudinal analyses of CT and tDCS effects. We will examine their effects on cognitive performance, functional and metabolic neuroimaging measures, and everyday functional abilities. At each assessment, we will obtain clinical and medical history, neurocognitive measures, and neuroimaging (structural MRI,

FMRI, MRS). All participants will undergo neuroimaging at baseline, following training, and at a three month follow-up.

## **Stimulated Brain Study**

| Screening | ✓ | ✓ | ✓ | ✓ | | | ✓ | | |
|---|---|---|---|---|---|---|---|---|---|
| Assessment<br>Visits 1-3<br>Activity<br>Summary | Informed<br>Consent<br>Form | Medical<br>History | Hearing<br>and Vision<br>Tests | Memory<br>and<br>Thinking<br>Tasks | Computerized Daily Activity Tasks, like banking etc. | Physical<br>and<br>Medical<br>Self<br>Reports | MRI<br>Screen-<br>Form | NIH tool<br>box | MRI<br>Brain<br>Scan<br>Appt. |
| Visit #1<br>Baseline | | | | ✓ | ✓ | ✓ | <b>√</b> | <b>√</b> | <b>√</b> |
| Visit #2 After 2 weeks (10 days) of Training | | | | <b>√</b> | <b>√</b> | <b>√</b> | ✓ | ✓ | ✓ |
| Visit #3 Three month followup | | | | <b>√</b> | <b>√</b> | <b>√</b> | ✓ | ✓ | ✓ |
| Daily Lab<br>Visits | Brain<br>Training<br>Games | Brain<br>Stimulati<br>on/Sham | tDCS<br>Sensation<br>Questions | | | | | | |
| Days 1-10 | ✓ | ✓ | ✓ | | | | | | |

- **6.2. Study participants and randomization procedure**. We will recruit 90 older adults (women = 45; age: 65-90 years). Study participants will consist of healthy individuals who have expressed an interest in taking part in an intervention aimed at optimizing and possibly preserving cognitive functioning and brain health. We will use web-based permuted block randomization to randomly divide participants into the four groups. People with pre-existing dementia, neurological brain disease, or meet criteria for a diagnosis of mild cognitive impairment (MCI) will be excluded, though people with subjective concerns about their cognitive functioning, who do not meet these criteria, may participate. Detailed inclusion/exclusion criteria can be found in Section 7.
- **6.2.1. Experimental Design Considerations and Limitations:** CT Approach. The POSITScience BrainHQ treatment program was selected because it 1) provides specific training tasks directed at three essential cognitive domains tied to our aims and hypotheses (attention, working memory, executive control) that correspond with the neurocognitive and functional neuroimaging measures to be studied; (2) is shown to produce significant cognitive and functional improvements with good effect sizes in past RCTs (ACTIVE) with up to 10 year durability and transfer of training to measures of self-reported everyday functioning; 3) provides a "cognitive treatment engine<sup>282</sup>" which alone has a very highly likelihood of yielding significant cognitive and functional improvements, enabling us to test the augmenting effects of tDCS; and 4) is computerized, well standardized, and efficiently implemented.

Combined CT. We selected a combined CT approach rather than testing one specific training task: 1) This would optimize CT treatment effects for this primary intervention, providing a strong and reliable engine of change with which to examine effects of tDCS; 2) This approach enables us to affect several related cognitive functions that are strongly dependent on neural plasticity of the frontal cortex; and 3) This approach would maximize participants interest and motivation versus a single task that could become boring.

<u>tDCS</u>. Brain stimulation provides a means of directly augmenting CT effects. tDCS was selected from possible alternatives (e.g., transcranial magnetic stimulation) based on research and data by Woods (PI), Hamilton, and Bikson (consultants), including its safety profile, ability to facilitate neural plasticity, and potential for application outside of research settings. Frontal stimulation was chosen based on prior and preliminary studies demonstrating significant impact on attention, working-memory, and other cognitive abilities to be trained during CT. 2mA tDCS was chosen based on prior research demonstrating that this parameter excites, rather than inhibits, activity in stimulated neurons. <sup>283</sup>

NIH Toolbox. A battery of neurocognitive tests was selected that could be completed in 1.5 hrs for all participants. A battery was selected that would enable optimal assessment of attention, executive functions, and working memory, but would also include some measures of learning and memory, and to a lesser extent other cognitive functions. We use the NIH Toolbox-Cognitive as a core element of this assessment, as it: 1) Can be completed in 30 minutes; 2) Is computerized and well standardized with norms from a large national cohort of older adults; 3) Provides both accuracy and response time measures; 4) Emphasizes the cognitive domains of relevance to the study; and 5) Has been the subject of considerable focus and investment by NIA. This study provides an ideal vehicle for implementing this battery. We supplement the Toolbox with measures to provide more coverage of working memory, attention, learning and memory.

# Stimulated Brain Surveys, Measures, Tasks and Activities Screening Visit:

#### **Informed Consent Process**

#### **Inclusion/Exclusion Screeners**

NACC UDS, Words in Noise (NIH-TB), Visual Acuity (NIH-TB), Colorblindness, MRI Screener, WTAR (optional: Mock MRI, MRI Measuring Device) Drug List review for inclusion/exclusion prescriptions

## **Baseline Computerized Tasks**

Posit Science Composite Baseline

#### **Psychological Measures**

BDI, Computer experience survey

## Demographic Information Medical History Form

## Assessment Visits: BL, POST, F/U

#### **Neurocognitive Assessment**

HVLT-R, STROOP, Trails A/B, BVMT-R, Digit Span, Timed Activities of Daily Living, COWA, PASAT, CALCAP

#### **Baseline Computerized Tasks**

Posit Science Baseline, NIH Toolbox, Functional Activities of Daily Living,

#### **Psychological Measures**

SF-36 Quality of Life, PSQ, STAI, BDI, AS, Computer experience survey, Expectations of brain training questionnaire, Expectations of brain stimulation questionnaire

#### **Physical Measures**

PROMIS Measure, tDCS Sensation Questionnaire, Grip Strength

## Mulitmodal Neuroimaging MRI Brain Scan

Baseline, Post, Three Month Follow-up

#### **Training Interventions:**

#### **Cognitive Training 5 hours per week**

(Posit Brain HQ 2 weeks)
Posit Baseline Measure/weekly

#### **tDCS Brain Stimulation**

(once per day for 10 days) tDCS Stimulation Survey/daily Electrode Drift Measurement

evaluation. All following assessments are identical otherwise.

Neuroimaging measures. We will focus on functional (FMRI) and cerebral metabolic (proton MRS) indices for two reasons: 1) These modalities are most linked to and likely sensitive to CT-associated neural plasticity and brain changes; and 2) Changes in these domains are likely to occur over the course of training compared to structural neuroimaging measures. We include active FMRI tasks related to the cognitive functions to be trained, as well as a passive resting state condition to examine the DMN. With respect to MRS, we use a single voxel method to achieve optimal sensitivity and will measure from two ROIs (frontal and posterior cingulate) corresponding to task and resting state associated brain areas. Along with Creatine (Cr), we will examine cerebral metabolites sensitive neuronal loss and membrane disturbances (NAA, GLx), and pro-inflammatory processes (Ch, MI). We will also measure cerebral GABA concentrations using a state of art MRS approach that will reflect neural plasticity in ROIs. The MRS indices will be examined for Aims 2. We will also collect FLAIR imaging data to assess white matter hyperintensity load, as a possible predictor of treatment response (secondary aim)

**6.3. Procedural sequence.** The sequence and flow of the assessments to be conducted at baseline and each subsequent assessment is shown below. We describe participant recruitment and retention strategies in the Human Subjects section. We will inform potential participants about the study, and obtain their consent. We will then screen for inclusion/exclusion criteria and schedule them for baseline assessment visit #1

**6.4 Cognitive Training.** CT will involve up to 10 hours of training over 2-weeks (10 days). At the screening visit, post 2-week intervention and the 3-month follow up visit, participants will complete a 20-minute composite measure of the cognitive training

tasks. <u>Training platform.</u> CT employs a PositScience BrainHQ suite via its researcher portal. These tasks are web-based and multi-platform (i.e., Windows, Mac). Participants will be randomly assigned to training on 4 tasks focusing on working memory or 4 tasks focusing on attention/speed of processing. Participants will be required to have a specific viewing distances. Study interventionists will provide daily performance summaries. The rationale and task demands for each component were described earlier (A.3.3). These CT are commercially available (<a href="https://www.positscience.com">www.positscience.com</a>), with well-documented protocols/manuals (See Appendix 1) and thus not described in detail here. (See miscellaneous attachments for specific game descriptions.) <a href="https://margiven.com/Hardware">Hardware</a>. Participants will complete CT on computers located at Clinical Translational Research Building. <a href="https://www.positscience.com">Support:</a> Participants will have the opportunity to ask questions, and will be instructed on the various computer tasks. No special technical skills or experience are required A support phone number will be available if participants have questions arise between study visits.

#### 6.5. Transcranial Direct Current Stimulation:

**Bilateral Frontal tDCS:** A Soterix Clinical Trials Direct Current Stimulator will apply 20 minutes of 2.0mA direct current through two biocarbon rubber electrodes encased in saline soaked  $5\text{cm}^2$  sponges (8cc of 0.9% saline solution) which then may be covered with electrode paste, and placed over the frontal cortices at F3 and F4 (10-20 system). Based on our well-established computational modeling workflow (C.4.1), F3/F4 stimulation delivers a broad pattern of frontal stimulation (see C.4.1d). Current inflow will occur on the right (F4), and outflow on the left (F3). Impedance quality will be ≤10kΩ to insure proper stimulation of brain tissue.

Sham tDCS: Sham stimulation is performed with the same device and all procedures will be identical except for the duration of stimulation. Participants will receive 30 seconds of 2 mA of direct current stimulation at the beginning of the session. Participants habituate to the sensation of tDCS within 30-60 seconds of stimulation. This procedure provides the same sensation of tDCS without the full duration of stimulation, making it a highly effective sham procedure. Blinding: The device has built in RCT double blinding protocols. Soterix will communicate only with Dr. Wu (Co-Mentor/statistician) to de-identify data for analyses.

<u>Physiological Recording</u>: During stimulation sessions participants will be asked to wear a special wristband that will be used to record physiological information such as pulse.

<u>3D Head Models of Electrode Placement and Electrode Drift Measurement:</u> We will take a brief set of images of the participant's head after the electrodes are placed to make sure that the electrodes are in the correct location. These images will be used to create a 3D model of the participant's head that will give us accurate information about where the electrodes were placed. In addition, we will physically measure any change in the electrode positioning over the course of the stimulation session to allow for assessment of quality control changes due to electrode drift. This is done by placing a mark at the bottom corners of each electrode and using a tape measure to measure the difference in electrode location at the end of the session. Ideally, no drift should occur and thus

measurement allows for use of a drift coefficient in statistical analyses of between participant differences in response.

6.6. Neuroimaging Methods. We will conduct neuroimaging on a Philips Achieva 3.0 Tesla research dedicated scanner with an existing research agreement. Scanning will take approximately 1 hour to acquire: 1) Structural MRI (T1, DTI), 2) FMRI (EPI-BOLD), 3) Proton MR Spectroscopy (MRS).

MRI Acclimation Protocol Options: Participants may have the MRI Measurement Tool (See MRI Measurement Tool Appendix in Misc. Attachments) demonstrated for them to visually see the size of the inside of the chamber of the MRI Scanner. Participants may be asked to try the device on themselves to gain a greater understanding of the size constraints related to the MRI Scan, and to give them a chance to experience the snug fit inside the core of the scanner. If participants cannot fit in the measurement device, they will be excluded from the study.

The participant may also be offered to make a visit to the Mock MRI Scanner (See Mock MRI Appendix in Misc. Attachments), located in the UF Dental Tower Ground floor, DG-73) to see if they are completely comfortable with the scanning process, and if they can realistically tolerate the size constraints. This can also be a time to discover if claustrophobia will be a limiting factor and exclusion for participation. If there is no concern regarding fit, or claustrophobia, this part may be skipped.

- **6.6.1. FMRI paradigms.** We will present the two FMRI tasks (2-Back, Spatial-Temporal Attention) using E-Prime 2 software (Psychology Software Tools, Inc., Pittsburgh, PA), with the video signal on a screen behind the participant's head. The screen is viewed through a double-mirror attached to the head coil. An MR-compatible piano-key response box attached to the stimulus presentation computer will collect performance data. We will apply a cushioned-pillow head stabilizer to minimize head movement during scanning.
- 2-Back. This task will measure brain changes due to our N-back training. We will assess verbal working memory on a 2-Back task, as in past studies 153,157. Consonants are visually presented for 500ms with an ISI=2500ms. Participants determine if each stimulus is the same or different from previously stimuli, responding by binary button press (yes vs. no). Executive control, phonemic buffering, and sub-vocal phonemic rehearsal are required. 0-back and 2-Back conditions are alternated in a block design with two 5-minute runs of eight blocks (consonant lists), with four blocks of the 0-Back and four blocks of the 2-Back. O-Back: Four blocks of nine consonants of random case and order (33% targets). Yes-no responses are made if targets that match stimuli occurring two earlier. 2-Back: Four blocks of 15 consonants (33% targets) will be pseudorandomly presented across the visual field. Accuracy and RT are recorded. The useful field of view (UFOV) fMRI task. Task will involve participants making decisions about where on the screen they saw a previously displayed object. Participants are presented two images simultaneously, one in a central box, and another outside the box. These images disappear very quickly and are replaced by a "noise" screen, similar to a scrambled television signal. Then participants are asked where they saw the object (a car) outside the box (e.g., up, down, left, right, etc.) and Protocol IRB #201400328 

what object was inside the box (either a car or a truck). The participants will respond using buttons on a response box. After participants have answered they are presented a fixation cross and wait until the next trial begins. Time between trials is randomized and jittered in accordance with best practice event-related fMRI design. The task duration is approximately 17 minutes. Examples of the stimuli are below.

## 1) Both objects are presented simultaneously



## 2) Noise Screen



**Resting State.** Participants will also be asked to rest for 6 minutes while functional data is being collected to assess resting state activation.

**6.6.2. Proton MRS:** GABA-edited spectra will be acquired using the MEGA-PRESS experiment, from 1 voxel (medial frontal). 9 minutes duration. Spectra will be analyzed using the Gannet package for the batch analysis of GABA-edited MR spectra, quantifying GABA concentration relative to water, correcting for voxel CSF fraction. OFF spectra will also be analyzed using LCModel to give concentrations for additional metabolites NAA, Glx, Cho, MI, and Cr. Analyses. Cerebral MRS metabolite concentrations will be derived from spectral analysis<sup>295</sup> With unsuppressed water FID at TE=30ms used for eddy-current correction. Time domain MRS ratios will be derived normalized for Cr. A double-exponential decay will be fitted to the water amplitudes at the 7 echo times. The signal amplitudes of brain tissue and CSF will be derived (corrected for T2 decay), with brain water signal used to correct for partial CSF volume. MRS Quality Assurance: GABA-edited MR spectra will be visually screened, and additionally spectra with a fitting residual of over 10% will be accepted for further analysis. The concentration measures for the additional metabolites will be accepted with an LCModel Cramer-Rao lower bounds (%SD) of less than 20%, a reliable estimate for a particular metabolite for group comparisons<sup>295</sup>. Scans resulting in spectra that do not meet quality criteria will be repeated. Past studies showed intra-subject variability of ~10% for GABA and 3-5% for other MRS peaks. Line width and signal-tonoise resonance ratios are plotted over time (brain, phantom) to monitor spectral

quality; inter- and intra-subject variability assessed by correlation and Bland and Altman plots. 412,413

- **6.6.3. Structural MRI.** High-resolution whole brain axial gradient-echo MPRAGE 3-D T1-weighted images will be acquired for volumetric and cortical thickness analyses and FMRI. <u>Analyses</u>: Volumetric indices will be obtained for total gray and white matter, FreeSurfer ROIs<sup>296-298</sup>, and a priori ROIs (MRS, FMRI).
- 6.6.4. **FLAIR**. Fluid attenuated inversion recovery (FLAIR) images will be acquired to assess white matter hyperintensity load (i.e., white matter damage). Volumetric and whole brain analyses of data will be used to look at region specific versus global levels of white matter load.
- 6.7. Neurocognitive and Psychological Assessments: Assessments will include a neurocognitive battery (approximately 180 minutes in duration, see list attached in Miscellaneous documents, and listed below. The battery consists of standardized, wellestablished neurocognitive measures with strong reliability and validity 304. Each is widely used in clinical neuropsychology and in Dr. Cohen's (Primary Mentor) research over the past 20 years. Our goal is to assess global cognitive ability (NIH-Toolbox: cognitive module), and specifically attention-executive functions, working memory, processing speed, and learning-memory. These are domains affected by aging<sup>24,31,146,305-314</sup> and will also tap the domains assessed by FMRI (Aim 1). Psychological measures are those commonly used in cognitive training paradigms, such as to gain greater understanding of the relation of things like depression, anxiety and apathy to the cognitive training intervention, and the resulting effect on memory and thinking. The BDI-II has a high risk of identifying severe depression and suicidality. The measure will be monitored carefully to identify and mitigate any risk to persons that are identified as at risk. The PI will be informed immediately, and a referral to Clinical and Health Psychology Clinic will be made right away for the participant. The PI or study staff will contact the participant directly to advise them of the concern, and assist with any intervention that may need to be referred. The State-Trait Anxiety Inventory(STAI) has medium risk to identify anxiety disorders and the same protocol will be followed if a participant is identified to have severe anxiety disorders that require medical treatment or referral to a Clinical and Health Psychology appointment for treatment. The National Alzheimer's Coordinating Center Uniform Data Set (NACC UDS), a comprehensive neuropsychological battery will be used to assess dementia/MCI in older adults. The NACC UDS is comprised of several neuropsychological tests including the Montreal Cognitive Assessment (MoCA), Craft Story Immediate and Delayed Recall (similar to the WMS Logical Memory), Benton Complex Figure Task Immediate and Delayed Recall, Number Span Forward and Backwards, Category Fluency, Trails A & B, The Multilingual Naming Test (similar to the Boston Naming Task), and Letter Fluency. The UDS takes approximately 45 minutes to administer. Score corrections are provided for age, sex and education.
- **6.7.1. Physical activity, QOL, PROMIS self-reported health assessment**. We will administer the, *Medical Outcomes Study Short Form-36 (SF-36: v.* 2.0, a widely used QOL measure), and the PROMIS self report measures at each assessment.

The PROMIS measures assess change in self-reported cognitive and physical function. <sup>321</sup> <sup>321</sup>. Change in self reported physical and mental health status correlate with QOL and mental and physical health status. <sup>322,323</sup> <sup>324</sup> These measures will serve as important assessments of interventions influence on everyday life.

## **Screening Visit**

Informed Consent

MRI Screener

Medical History/Prescription Drugs

**Drug Exclusion List Review** 

**NACC UDS** 

Words in Noise (NIH-TB), Visual Acuity (NIH-TB), Color Vision

WTAR

Posit Composite Baseline Game Testing (0%-79% range)

BDI

Computer and Technology Use Questionnaire

## Assessment Visits #1,2,3

NIH Toolbox

**HVLT-R** 

**BVMT** 

Stroop Test

Trails A & B

**COWA** 

**Apathy Scale** 

SF 36 Quality of Life

PROMIS self-report

Digit Span

Pittsburgh Sleep Questionnaire

Pain Questionnaire

BDI/STAI

**PASAT** 

**CALCAP** 

Expectation of brain stimulation questionnaire

Expectation of brain training questionnaire

## Daily Check In

tDCS Stimulation sensation questionnaire

#### 7. Possible Discomforts and Risks:

#### Potential Risks.

There are minimal risks associated with participation in this study. The potential risks are as follows:

Magnetic resonance imaging (MRI). MRI is a procedure that allows doctors to look inside the body by using a scanner that sends out a strong magnetic field and radio

Protocol IRB #201400328


waves. This procedure is used routinely for medical care and is very safe for most people, but you will be monitored during the entire MRI scan in case any problems occur. The risks of MRI as detailed in the Informed Consent are:

- The MRI scanner contains a very strong magnet. Therefore, you may not be
  able to have the MRI if you have any type of metal implanted in your body, for
  example, any pacing device (such as a heart pacer), any metal in your eyes, or
  certain types of heart valves or brain aneurysm clips. Someone will ask you
  questions about this before you have the MRI.
- There is not much room inside the MRI scanner. You may be uncomfortable if you do not like to be in close spaces ("claustrophobia"). During the procedure, you will be able to talk with the MRI staff through a speaker system, and, in the event of an emergency, you can tell them to stop the scan
- The MRI scanner produces a loud hammering noise, which has produced hearing loss in a very small number of patients. You will be given earplugs to reduce this risk, and headphones for added protection.
- If you are a woman of childbearing potential, there may be unknown risks to the fetus. Therefore, before you can have the MRI, you must have a pregnancy test.
- If an obvious abnormality is discovered during your MRI scan, you will be informed about it by the research team, you will be provided with a copy of your MRI scan and we will encourage you to see your primary care physician. MRI will only be done for research purposes in this study.
- You will be monitored very carefully while in the scanner, and repeatedly checked to ensure comfort.

There is a risk of introducing metal into an MRI environment. However, the MRI compatible transcranial direct current stimulator contains no materials that respond to the MRI environment. Thus, the risks associated with undergoing MRI while receiving stimulation are the same as transcranial electrical stimulation outside the MRI scanner.

<u>Transcranial direct current stimulation.</u> Transcranial direct current stimulation is considered safe but a small number of people do experience some side effects. The most common side effects are itching and tingling or mild discomfort at the area of stimulation, and headache. Other possible side effects include dizziness and nausea. Whenever an electrical stimulation is applied to the body, it could possibly cause a seizure or abnormal heartbeat, but this has never occurred with the transcranial direct current stimulation parameters used in this study.

Although there is no known risk to pregnancy, there may be unknown risks and all women of child bearing potential must have a negative pregnancy test prior to stimulation.

<u>Cognitive Training.</u> There is a risk participants will find cognitive training on the computer challenging, fatiguing, and/or boring. Research staff will explain what to do and how to perform the training tasks tests during your initial study visit. Participants will also have access to a 24-hour help line should you have trouble working with the training computer.

<u>Neurocognitive and Functional tests</u>. There is a risk that you will find cognitive and functional tests challenging, because it may be difficult to remember the things that you are asked to remember or have trouble hearing or seeing some of the sounds and pictures presented on the computer screen. You may skip any tests you do not wish to complete. Research staff will explain what to do and help you take the tests during your study visit.

<u>Questionnaires</u>. There is a risk that you will find questions on the questionnaires uncomfortable to answer. You may skip any question you feel uncomfortable answering.

Other possible risks to you may include fatigue due to the testing. Should this occur, you can take a rest-break at any time or you may discontinue the testing at any time. If requested by the participant, multiple test days are possible.

When being tested some people may develop anxiety. If these tests make you anxious we can stop the testing.

Researchers will take appropriate steps to protect any information they collect about you. However, there is a slight risk that information about you could be revealed inappropriately or accidentally. Depending on the nature of the information, such a release could upset or embarrass you, or possibly affect your insurability or employability. Questions 17-21 in this form discuss what information about you will be collected, used, protected, and shared.

This study may include risks that are unknown at this time.

Participation in more than one research study or project may further increase the risks to you. If you are already enrolled in another research study, please inform one of the research team members listed in question 3 of this form or the person reviewing this consent with you before enrolling in this or any other research study or project. If you are currently participating in another study using transcranial direct current stimulation or transcranial magnetic stimulation, you will be rescheduled so that your participation in the current study does not overlap with your participation in the other study.

## Adequacy of Protection against Risks.

Recruitment and Informed Consent. All study participants will provide written informed consent. Persons will be recruited from the CAM-CTRP research registry, community outreach, or community agencies. Participants will also be recruited at community events with IRB-approved flyers, and participants will have the option to confidentially provide name, phone number, and email if they wish to be contacted by the study team to determine study eligibility. The contact information will be securely stored during the

event and immediately stored in the Woods Lab per study data safety management plan. People interested in participating in the study will call the CAM-CTRP study recruitment coordinator. Potential participants interested in hearing more about the study will be provided information about the study. Persons will then indicate their agreement to participate by signing the informed consent document.

Our inclusion and exclusion criteria are designed to minimize risks to participants.

*Inclusion criteria*: 1) Men and women; 2) Age: 65 to 90 years; 3) English speaking; 4) Physically mobile; 5) working memory function between 0-75<sup>th</sup> percentile determined by screening results on the POSIT Baseline Cognitive Training computerized tasks.

Rationale: (1) The age range is selected to include a higher proportion of persons with possible concern about cognitive deficits (2) The language requirement will avoid difficulties with interpretation of cognitive results; (3) the mobility requirement is required because participants will need to be able to participate in neurocognitive testing and MRI testing at different locations; 4) the working memory function requirement is needed to avoid randomized groups from being biased by over-representation of extremely high (e.g., super agers) working memory function in a particular group and to include a representative sample consistent with the "typical" cognitive aging profile in US.

**Exclusion criteria**: 1) Neurological disorders (e.g., dementia, stroke, seizures, traumatic brain injury). 2) Evidence of dementia (NACC UDS scores of 1.5 standard deviations below the mean for age, sex and education adjusted norms in a single cognitive domain on the task). 3) Past opportunistic brain infection 4) Major psychiatric illness (schizophrenia, intractable affective disorder, current substance dependence diagnosis or severe major depression and/or suicidality. 5) Unstable (e.g., cancer other than basal cell skin) and chronic (e.g., severe diabetes) medical conditions. 6) MRI contraindications (e.g., pregnancy, claustrophobia, metal implants that are contraindicated for MRI). 7) Physical impairment precluding motor response or lying still for 1 hr and inability to walk two blocks without stopping.8) Certain prescription medications may possibly reduce effects otherwise induced by the tDCS stimulation protocol, and are listed on a Drug Exclusion List attached to the Appendices in Miscellaneous attachments of this study. 9) Hearing or vision deficits that will not allow for standardized cognitive training stimulation; ie colorblindness, inability to hear through headphones (with or without hearing aids), macular degeration or other significant diseases that cause severe loss of vision. If vision is corrected with lenses to appropriate levels, then participant will be eligible. 10) Left handedness, as those with left-handedness have a higher percentage rate of atypical functional lateralization for brain functions, which would significantly interfere with interpretability of brain data.

Rationale: (1) neurological diseases affecting the brain create obvious confounds that would obscure the study's findings or increase risk from non-invasive brain stimulation (i.e., seizures). (2) The NACC UDS will be used to exclude people meeting criteria for severe dementia, as this study is focused on more mild cognitive deficits; (3) past opportunistic brain infection, and (4) a history of severe psychiatric illness

(schizophrenia, chronic intractable unipolar or bipolar depression) also would directly affect neurocognitive test performance and thus would confound study findings. (5) Unstable (e.g., cancer) and certain chronic medical conditions (e.g., severe obesity) may also confound findings and increase study attrition; (6) Given that this study requires MRI imaging to address all aims, factors that make MRI imaging unsafe or infeasible for particular study candidates will serve as a basis for exclusion; and (7) Physical limitations are a basis for exclusion based on inability to participate in all study procedures. Excluding people who cannot walk or sit for an hour will reduce problems in the scanner that could confound study findings.

## Protection against Risk.

Protection against Risk of confidentiality. Information pertaining to research subjects will be obtained from (1) interviews with subjects and (2) procedures described in the "research design and methods" section. All data will be considered confidential according to HIPPA guidelines for personal health information. All participants will sign a combined consent to participate in research and HIPPA compliant confidentiality document approved by the IRB overseeing the clinical recruitment setting (i.e. the University of Florida IRB, and the Florida Department of Health IRB).

Precautions will be taken to ensure that all research materials are inaccessible to anyone other than the investigators, and by ensuring that only qualified and trained individuals conduct the study research procedures. Prior to study initiation, procedures for protecting the confidential nature of participant data collected will be reviewed and all questions or concerns will be clarified at this time. These procedures will be reviewed throughout the study. Staff will be trained and certified in handling human subject information to maintain privacy and confidentiality. Procedures for allowing access to investigators to use this information for research will be under the authority of the PI and will follow HIPPA compliant guidelines for the release of PHI.

Contact information for study participants will be kept in separate files and databases from the research data. This information will be used by the research assistants to send reminders about follow-up times and appointments via phone, email or mail correspondence. The information will only be kept on computers or devices that are both password protected and encrypted. Any written forms will be kept in locked file cabinets or locked briefcases. None of the research data in the central data base will have participant identity information. No results will ever be reported in a personally identifiable manner. All research data will be entered directly into a web-based survey that is maintained by the University of Florida CTSI (REDCap), and the data are encrypted as soon as they are sent in a wireless format. The data will be transferred and stored on secure servers at the University of Florida, with no identifying information.

No survey data will be labeled with the participant's name or other identifying information, but will instead be labeled with a study ID number. Documents linking study ID numbers to identifying information (e.g., name, address, etc) will be stored electronically in a password-protected file. All paper-data with identifying information will be stored in locked file drawers, separate from coded data. Documents linking study ID

numbers to identifying information will be destroyed at the end of the study. Documents containing data collected on un-consented individuals (i.e., screening logs used to avoid approaching the same individual for study enrollment twice) will be shredded daily. All electronic data will be secured and encrypted. Identifying information will not be reported.

*Protections of risks related to study questionnaires*. To minimize any risks related to emotional responses to questionnaires, persons will be informed about the types of questions included in the surveys, which are similar to the types of questions persons might be asked by their doctor in a clinical setting.

Protection of risks related to tDCS. To minimize risk associated with tDCS, participants will be monitored throughout stimulation sessions and asked to report any discomfort. If scalp sensation is uncomfortable, stimulation levels will be decreased to a comfortable level or will be stopped. In the event of a headache, stimulation will be decreased to a comfortable level (where the headache or nausea is no longer present) or will be stopped. All tDCS sessions will be administered and continually supervise by a trained experimenter. The above symptoms have only been reported when participants are actively being stimulated. However, to assess for any symptoms occurring during the 24 hour interval between stimulation sessions, we will administer a brief symptom screening questionnaire at the beginning (symptoms in the past 24 hours) and end of each session (symptoms during stimulation). tDCS has not been shown to cause seizures nor lower the seizure threshold in animals. There are no reports of seizure induced by tDCS in human participants in the literature. However, this may not be true for epilepsy patients, whose seizure threshold rates are likely abnormal. Prior history of neurological disorders is an exclusionary criterion for our study and thus no participants will have a history of seizure.

Protection against risks associated with neuroimaging. MRI is widely regarded as a safe, noninvasive procedure for visualization of brain tissue in both adults and children. Prior fMRI studies by our group and by other groups document the innocuous nature of these procedures. Prior to study participation, all participants will be informed of the MRI procedure during the informed consent/assent process. The proposed study will be performed on an FDA approved Phillips 3 Tesla scanner located at the Advanced Magnetic Resonance Imaging and Spectroscopy (AMRIS) research facility at UF. There are no known long-term effects of MRI procedures on the body. The FDA Information Sheets, Food and Drug Administration, October 1995, p. 79, lists as a non-significant risk device, "Magnetic Resonance Imaging (MRI) Devices within FDA-specified parameters." This study satisfies those parameters. The 3.0 tesla MR scanners meets FDA parameters for field strength, gradient switching, and RF power deposition for all FDA-approved acquisition schemes including echo-planar imaging. In addition, this research protocol involves the use of an FDA-approved acquisition scheme, or the power deposition of experimental acquisition scheme proposed meets FDA parameters as verified on a phantom using the power monitoring system installed on the MR scanner. Both Dr. Woods and trained MRI staff will check for exclusion criteria. The main MRI-related risks include: (a) sensitivity to the loudness of the MRI machine - all subjects will be given and must wear ear plugs; a squeeze-ball and microphone will be

provided so that they may stop the testing if they become uncomfortable or anxious at any time; (b) claustrophobia - subjects will have the opportunity to practice in a simulator and to become as familiar and comfortable as possible before commencing the experiment. In addition, they will be given the opportunity to examine the scanner before the tasks starts. The study will be ended early if the space is a problem for them: no medications (e.g., benzodiazepines or tranquilizers) will be offered to them; (c) lightheadedness when sitting up after lying in the MRI machine - this feeling sometimes occurs but has always gone away in a few minutes. Participants will thus be assisted in getting up to make sure they do not fall; (d) risks associated with having an MRI in pregnant women - while risks to pregnant women have not been conclusively documented, reports of potential risk to unborn fetuses have prompted the exclusion of these individuals from research. Given the age range of our sample, the probability that one of our female subjects will be pregnant is relatively low. Nevertheless, as a standard procedure, all female participants will undergo a test to determine pregnancy prior to entering the MRI. In sum, the MRI neuroimaging procedures pose no radiological or medical risk, given that participants with metal implants susceptible to magnetic heating will be excluded based on standard scanner policies. A small number of people may become anxious in the small space of the scanner. These individuals will have the opportunity to terminate the scan session. Furthermore, all recruits will be screened for phobias prior to enrollment. FMRI procedures will be supervised by Dr. Woods, a close collaborator with Dr. Song Lai, the MR physicist in charge of the facility. There is a medical technologist at the imaging site at all times to insure scanner safety, and neuroradiologists on call as needed. If an abnormality is noted on the structural MRIs by study staff, the PI will provide the participant with a copy of the scan and encourage them to follow up with a neurologist.

Protection against risks associated with neurocognitive tests. The neurocognitive assessments have minimal risk associated with them. Some participants experience stress associated with being tested, though this tends to be quite limited. Breaks will be given in those cases. Research staff that collect data have been trained in the conduct of all cognitive function tests by other senior staff members. Research staff members will be certified in the conduct of the cognitive function tests before they work with study participants.

## **Data and Safety Monitoring Plan:**

A data and safety monitoring plan (DSMP) will be implemented to ensure the safety of all participants involved in the study and to ensure the validity and integrity of the data. The PI will be responsible for coordinating activities of the DSMP, including: arranging meetings and communications, and identifying and reviewing relevant participant materials. The data and safety information obtained on each study participant will be reviewed at weekly meetings. The primary goal of the DSMP will be to monitor the progress of the study and safety of participants and if necessary, recommend modifying the study or terminating the study as appropriate.

Concerns that might dictate modification or termination of the study include:

- Participant safety
- Outcome data
- Data quality
- Integrity
- Intervention efficacy
- Recruitment
- Performance

Both the PI and the study staff will review the study weekly and examine reports of adverse incidents and reports of study participant recruitment and follow-up. Throughout the course of the study, information regarding issues deemed critical to the study or to the safety of research participants will be provided to the PI and primary mentors. As a result of receiving this critical information, a meeting to discuss this information may be convened. Information deemed critical would include:

- Serious and non-serious adverse events that may occur
- Suspicion of scientific fraud or misconduct
- Any other issues which may warrant protocol changes or modifications.

Because this is an exploratory study with minimal risk associated with the proposed intervention and limited financial resources, there will not be an external data safety and monitoring board for this study. The research team, however, will follow the procedures for data safety and monitoring as required by the Institutional Review Board at the University of Florida (UF IRB).

The research team will monitor participants for any potential adverse events, and all reported events will be forwarded by the PI to the UF IRB.

Procedure for collection and storage of data. A number of quality control procedures will be used to ensure the validity and integrity of the data and the safety of all participants involved in the study. Relevant data and safety information obtained on each study participant will be verified against the original source documents by the primary study coordinator and any identified discrepancies will be reviewed at these weekly meetings. The primary goal of these meetings will be to monitor the progress of the study and safety of participants and if necessary, recommend modifying the study or terminating the study as appropriate.

All identifying information will be archived in Dr. Woods' neuroimaging laboratory within the Center for Cognitive Aging and Memory at UF. Imaging data will undergo several levels of processing, and all raw and processed data will be archived on a password-protected server in password-protected folders and files. Only study staff will have access to these files. The self-report data will be double entered using the SPSS Data Entry system. This system signals the user when an out-of-range value is entered. All data entry is then verified via double-entry, with the program signaling mismatches with the original entry. Next, computer-generated reports of variable frequencies and subject lists will be reviewed, leading to possible corrections to coding or entry. After checking for accuracy of data within a given group, data will be stored in the password-protected folders along with the imaging data.

Location and logistics of data collection. All procedures involving human subjects will be performed at facilities of the UF Health Care System. Neurocognitive testing and training will be performed at either the Clinical and Translational Research Institute or the AMRIS/MBI UF facility. Several clinical research examination rooms are equipped and dedicated to neurocognitive and functional assessment, and contain all necessary computers and test materials. Blood for serum biomarker analysis will also be collected at this site. The Clinical and Translational Research Institute (CTSI) which contains laboratories, freezers, and main frame computers. Storage of neuroimaging data backup will occur there. Neuroimaging will take place at the AMRIS facility of the McKnight Brain Institute.

Storage of collected data. All electronic data are stored in password protected, secured computer systems. All paper data will be stored in a locked file cabinet. Data will only be removed when coded, entered, or audited. Only the participant's study identification number will appear on any data forms. Only the PI, the Co-Is, and the RAs will have access to the completed data forms and electronically stored data. All data are considered part of the participant's confidential record. Data collected from research participants will be stored in a secured, password protected computer file that is separate from network systems. All paper data (e.g., subject contact information, consent forms, etc.) will be placed in a locked file cabinet within 24 hours of their acquisition as designated by the study's RA. All data will remain confidential. A file will be maintained that associates the participant's name with that participant's study identification number. This file will be kept in a locked cabinet separate from the study data

Data entry requirements. The data entry system will require a login identification and password in order to gain access to the data. Where appropriate, validation and range rules will be applied to the actual entry fields. Only the PI and Co-Is will be able to view the data in its raw state.

Audit/verification of entered data. All data designated as primary outcome data will be subject to a 100% cross-referencing between electronic and paper forms. This audit must have an error rate less than 1%. If the verification fails the audit, all data will be reentered, the original computer files discarded, and the newly re-entered data audited. This process will continue until the audit no longer exceeds the maximum allowable error rate. All audits will be supervised and documented by the PI.

Data management and analysis. Our research team has substantial experience in the design and implementation of data management procedures that provide accurate recording and storage of data, participant confidentiality, and timely analysis. Based on our past experience, we believe that our major data management and analysis needs for the proposed project can be met by using a high-end PC, equipped with the latest version of SPSS for Windows and appropriate spreadsheet programs. All data files are automatically backed-up daily.

Data quality control. All staff involved in data collection will be trained and certified to ensure their competence, and re-certified periodically throughout the study as we have done in similar trials. Data will be collected and numerically coded using pre-tested electronic entry forms. At the time of collection, there will be initial clerical review of all Protocol IRB #201400328  data for accuracy and completeness. Every effort will be made to ensure that missing data are kept to a minimum. Data entry programs with range checking and response validation will be used for all data entered. Under supervision from the PI, the data manager will conduct error checking procedures and preliminary analyses on all data to ensure their accuracy. The RAs will be trained to avoid omissions in data entry and computer entry protocols will be programmed to avoid accidental skipping of question items. We believe that the quality control system to be used will ensure a complete and accurate database, and maximize the likelihood that the intervention will be delivered correctly and efficiently. As we have done in prior studies, a manual of procedures will be developed during the initial study start-up period that explicitly describes the specific procedures related to intervention delivery, data collection, and quality assurance.

<u>Frequency of data review.</u> Relevant data and safety information obtained on each study participant will be verified against the original source documents by the primary study coordinator on a bi-weekly basis. As noted above, any identified discrepancies will be discussed with the Principal Investigator and reviewed at weekly meetings.

Measurement and reporting of participant accrual and adherence to eligibility criteria. Review of the rate of participant accrual, adherence to inclusion/exclusion criteria will occur weekly during the recruitment phase and then every month to assure that participants meet eligibility criteria and ethnic diversity goals outlined in the grant proposal.

<u>Designation of an independent monitoring committee</u>. The Independent Monitoring Committee for this study will consist of an established board which has reviewed all studies conducted within the CAM-CTRP during bi-annual conference calls for the past six years.

Safety Review Plan Study progress and safety will be reviewed monthly (and more frequently if needed) by the principal investigator. Progress reports, including participant recruitment, retention/attrition, and AEs will be provided the IoA Independent Monitoring committee for bi-annual reviews. An annual report will be compiled and will include a list and summary of AEs. In addition, the annual report will address (1) whether adverse event rates are consistent with pre-study assumptions; (2) reason for dropouts from the study; (3) whether all participants met entry criteria; (4) whether continuation of the study is justified on the basis that additional data are needed to accomplish the stated aims of the study; and (5) conditions whereby the study might be terminated prematurely. The annual report will be signed by the chair of the Independent Monitoring Committee and may be forwarded to the IRB, NIH, & CTSI. The IRB and other applicable recipients will review progress of this study annually.

<u>Final storage of paper data.</u> All paper data (e.g., consent forms) will be housed at a facility that specializes in the storage of medical/ research information. The destruction date of these files will be at least 7 years from the termination of the study and will be authorized by the Principal Investigator of the research study.

Access to cleaned computer data. Once the study is complete, and all data have been collected, entered and passed the audit process, the data will be available to the Principal Investigator and his designates for analysis. Only the Principal Investigator can

give permission for the release of aggregated study data. No confidential information may be released without the express written consent of the study participants. Only copies of the finalized data will be released. The original data file will remain in its pristine state.

Monitoring physical health and safety. All assessment visits will be conducted at a central location and all testing sessions will be conducted and supervised by a trained and certified research staff that will monitor potential adverse experiences and symptoms. At each visit, participants will be asked to report any adverse events they have experienced since their last visit. Immediate medical treatment will be provided for any illness or injury resulting from this study. Trained nursing staff members are present in the research center at all times, and a physician will also be available to evaluate the participant if needed.

In addition to the assessments conducted at in-person study visits, participants will be contacted by phone on a <u>weekly basis</u> between the end of training and the 12-week follow-up visit and will be asked to report any adverse events that have occurred since their previous phone contact or study visit. Specifically, they will be asked about any adverse events, including itching, pain, nausea, headache, etc. they have had. Participants will also be asked about their mood, including depressive symptomatology, and other health related activities (i.e., physical activity), as well as general health status. Based on reported symptoms, participants may be asked to come in for an additional follow-up assessment visit with one of the healthcare professionals on the study team (i.e., physician or psychologist) for further evaluation of their symptoms. Based on information obtained at this visit, participants will then be referred for follow-up assessment and/or treatment with the appropriate healthcare provider.

Monitoring mental health and safety. At each assessment visit, participants will complete the BDI to assess for depressive symptom severity. Any participant who endorses clinical levels of any psychiatric disorder or who endorses suicidality will be referred to Dr. Cohen, study psychologist, for further follow-up assessment. The psychologist will then provide a recommendation regarding the appropriate course of follow-up and also advise on whether it is safe for the participant to continue in the study. If a participant is found to be actively suicidal with a plan and/or intent, they will be escorted immediately to the emergency room at the Shands Hospital at the University of Florida. If safety is an issue, UF security or local authorities will be called for assistance. If a participant endorses suicidal thoughts or significant psychopathology, participants will be referred for further by evaluation with Dr. Whitehead (Licensed psychologist and co-investigator). Based on this evaluation, she will recommend follow-up assessment and treatment appropriate to the situation including treatment at the Psychology and/or Psychiatry Clinics within Shands Hospital at the University of Florida.

<u>Adverse Event Reporting.</u> An adverse event (AE) is defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the intervention irrespective of whether it is considered related to the intervention.

Non serious adverse events. Defined as conditions that may be unpleasant and bothersome to the participant that does not require discontinuing the study.

Serious adverse events (SAEs). Defined as events that may be harmful to the participant and/or may be serious enough to warrant either temporary or permanent discontinuation of the study intervention, either because they are intolerable or because they are judged to be potentially harmful. All serious adverse events require immediate reporting and an assessment of the implications for the continuation of the study and/or modification of the consent form. The following are considered serious events:

It is acute or life threatening;

It results in prolonged, permanent or severe disability;

It is another severe illness including worsening of a pre-existing condition, injury or accidents;

It is an inpatient hospitalization or surgical procedure, or a treatment to prevent a serious event:

It results in death:

It is a clinically significant abnormal laboratory or diagnostic test.

Table 3. Adverse Event (AE) Classification

| Adverse Event (AE) Classification | |
|---|---|
| Definite. | Temporal pattern + known or expected AE response pattern + confirmed by |
| | stopping the intervention + reappearance of AE on re-challenge |
| Probable. | Temporal pattern + known or expected AE response pattern + confirmed by |
| | stopping the intervention + could not be explained by participant's clinical |
| | state |
| Possible. | Temporal pattern + known or expected AE response pattern + could have |
| | been produced by a number of other factors |
| Unknown. | Relationship for which no evaluation can be made |
| Not related. | AE for which sufficient information exists to indicate that the cause is |
| | unrelated to the study intervention |

Classification of AE severity. The principal investigator will

evaluate adverse events for seriousness, expectedness, severity, and relationship to study intervention at each study visit. The primary mechanism for ensuring participant safety will be clinical observation of symptoms. The study will be conducted and supervised by trained study staff that are certified in CPR and will monitor potential adverse experiences and symptoms. During each visit, participants will log any healthrelated problems or symptoms they are experiencing. These sheets will be reviewed by study staff before allowing the participant to continue. Community health services will be contacted immediately if warranted by the participants' symptoms.

All adverse events (AEs) will also be categorized according to the likelihood that they are related to the study intervention. Specifically, they will be labeled either definitely, probably, possibly or unrelated to the study intervention. The classification of potential relationship to the intervention is shown in Table 3.

Effective screening will exclude individuals who would be at increased medical risk as a result of participation in this research. FMRI contraindications, such as claustrophobia or some metal implants will be assessed by telephone screening and again on the day of the scan. Dr. Woods, who has completed MRI safety training and Protocol IRB #201400328  has over 4 years experience screening FMRI participants, will supervise these procedures. The RA who will conduct neuroimaging analyses will be trained in UF AMRIS safety procedures and will also be responsible insuring for participant safety. Adverse events, although unlikely, may occur as a result of neuroimaging. Such events will immediately be reported by Dr. Woods (PI) to the local IRB, with serious adverse events reported to both the IRB and NIH.

<u>SAE reporting.</u> Serious adverse events (SAEs) that are unanticipated, serious, and possibly related to the study intervention will be reported within 24 hours of study's knowledge of the SAE to the Independent Monitor, IRB, and CTSA in accordance with the regulatory requirements. Anticipated SAEs or those unrelated to the study intervention will be reported to the same individuals/entities in accordance with regulatory requirements.

Minor events will be reported to the IRB at the time of annual review, as well as to the oversight committee on a bi-annual basis. Both the principal investigator and the study staff will review the study weekly and examine reports of adverse incidents and reports of study participant recruitment and follow-up. Throughout the course of the study, information regarding issues deemed critical to the study or to the safety of research participants will be provided to the principal investigator and other study investigators as needed. As a result of receiving this critical information, a meeting to discuss this information may be convened. Information deemed critical would include:

- serious and non-serious adverse events that may occur;
- · suspicion of scientific fraud or misconduct;
- any other issues which may warrant protocol changes or modifications.

Adverse event (AE) and serious adverse event (SAE) determination and monitoring will be achieved via administration of structured questionnaires. Standardized forms for referring and treating study participants who experience adverse events will be in place.

<u>Documentation of Training on Protection of Human Participants.</u> All key personnel on the study have successfully completed and obtained certification from their respective institutions for Mandatory Education in Human Research Subjects Protection. The Mandatory Education is described as follows:

On August 23, 2000, an institutional policy was enacted requiring all clinical investigators and their key personnel to undergo mandatory education in human research subject protection. The program was initiated on September 1, 2000 and includes all clinical researchers regardless of source of research funding. At the core of the self-directed training program is the tutorial manual entitled, "Protecting Study Volunteers in Research" by Dunn and Chadwick. Each researcher receives a copy of the manual and, in a timely fashion, completes the test included in the manual. Each researcher must obtain a score of >86 to complete the certification requirements to conduct clinical research at this institution. In all cases, no researcher will be allowed to conduct clinical research without proof of human research subject protection education after September 30, 2001.

Additional and continuing education opportunities for clinical researchers include the Office of Research Administration newsletter that is circulated to approximately 900 recipients every 6 weeks. Relevant information concerning research review is available on the UF ORA web page. In addition to standard institutional research information, the web page contains links to other sites such as CenterWatch, NIH.

## 8. Possible Benefits:

There are well-documented benefits for older adults who participate in cognitive training, including improvement in working memory, attention, and executive functions. Deficits in these cognitive abilities significantly impact quality of life, financial capacity, medication adherence, and mortality in older adults. All participants undergoing CT may benefit from these effects. Those participants randomly assigned to the active tDCS+CT treatment group may experience further benefit beyond that of cognitive training alone. Benefits to society will include the contribution of novel data regarding the efficacy of neuromodulation methods for enhancing cognitive training effects in older adults. This may help inform treatment protocols in a growing segment of the US population (i.e., those 65 years and older). Data collected from this study will serve as a foundation for larger clinical studies that examine optimized methods for treating aging-related cognitive decline using cognitive training and tDCS. Some participants may not benefit from the study at all.

#### 9. Conflict of Interest:

None

#### References:

- 1. Sumner P, Edden RA, Bompas A, Evans CJ, Singh KD. More GABA, less distraction: a neurochemical predictor of motor decision speed. *Nat Neurosci.* Jul 2010;13(7):825-827.
- 2. Streeter CC, Jensen JE, Perlmutter RM, et al. Yoga Asana sessions increase brain GABA levels: a pilot study. *J Altern Complement Med.* May 2007;13(4):419-426.
- 3. Edden RA, Muthukumaraswamy SD, Freeman TC, Singh KD. Orientation discrimination performance is predicted by GABA concentration and gamma oscillation frequency in human primary visual cortex. *J Neurosci*. Dec 16 2009;29(50):15721-15726.
- 4. Puts NA, Edden RA, Evans CJ, McGlone F, McGonigle DJ. Regionally specific human GABA concentration correlates with tactile discrimination thresholds. *J Neurosci.* Nov 16 2011;31(46):16556-16560.
- 5. Gao F, Edden RA, Li M, et al. Edited magnetic resonance spectroscopy detects an age-related decline in brain GABA levels. *Neuroimage*. Sep 2013;78:75-82.
- 6. Streeter CC, Whitfield TH, Owen L, et al. Effects of yoga versus walking on mood, anxiety, and brain GABA levels: a randomized controlled MRS study. *J Altern Complement Med.* Nov 2010;16(11):1145-1152.

- 7. Cohen RA, Moser DJ, Clark MM, et al. Neurocognitive functioning and improvement in quality of life following participation in cardiac rehabilitation. *Am J Cardiol.* May 1 1999;83(9):1374-1378.
- 8. Osowiecki DM, Cohen RA, Morrow KM, et al. Neurocognitive and psychological contributions to quality of life in HIV-1-infected women. *AIDS*. Jul 7 2000;14(10):1327-1332.
- 9. Al-Khindi T, Macdonald RL, Schweizer TA. Cognitive and functional outcome after aneurysmal subarachnoid hemorrhage. *Stroke; a journal of cerebral circulation*. Aug;41(8):e519-536.
- 10. Wadley VG, Crowe M, Marsiske M, et al. Changes in everyday function in individuals with psychometrically defined mild cognitive impairment in the Advanced Cognitive Training for Independent and Vital Elderly Study. *J Am Geriatr Soc.* Aug 2007;55(8):1192-1198.
- 11. Soderqvist A, Miedel R, Ponzer S, Tidermark J. The influence of cognitive function on outcome after a hip fracture. *The Journal of bone and joint surgery*. Oct 2006;88(10):2115-2123.
- 12. Ettenhofer ML, Hinkin CH, Castellon SA, et al. Aging, neurocognition, and medication adherence in HIV infection. *Am J Geriatr Psychiatry*. Apr 2009;17(4):281-290.
- 13. Ochner CN, Green D, van Steenburgh JJ, Kounios J, Lowe MR. Asymmetric prefrontal cortex activation in relation to markers of overeating in obese humans. *Appetite*. Aug 2009;53(1):44-49.
- 14. Reijnders J, van Heugten C, van Boxtel M. Cognitive interventions in healthy older adults and people with mild cognitive impairment: a systematic review. *Ageing Res Rev.* Jan 2013;12(1):263-275.
- 15. Li H, Li J, Li N, Li B, Wang P, Zhou T. Cognitive intervention for persons with mild cognitive impairment: A meta-analysis. *Ageing Res Rev.* Apr 2011;10(2):285-296.
- 16. Papp KV, Walsh SJ, Snyder PJ. Immediate and delayed effects of cognitive interventions in healthy elderly: a review of current literature and future directions. *Alzheimers Dement*. Jan 2009;5(1):50-60.
- 17. Ball K, Edwards JD, Ross LA. The impact of speed of processing training on cognitive and everyday functions. *The journals of gerontology. Series B, Psychological sciences and social sciences.* Jun 2007;62 Spec No 1:19-31.
- 18. Cicerone KD, Dahlberg C, Kalmar K, et al. Evidence-based cognitive rehabilitation: recommendations for clinical practice. *Arch Phys Med Rehabil.* Dec 2000;81(12):1596-1615.
- 19. Ball KK, Beard BL, Roenker DL, Miller RL, Griggs DS. Age and visual search: expanding the useful field of view. *Journal of the Optical Society of America. A, Optics and image science.* Dec 1988;5(12):2210-2219.
- 20. Ball K, Owsley C. The useful field of view test: a new technique for evaluating age-related declines in visual function. *Journal of the American Optometric Association*. Jan 1993;64(1):71-79.
- 21. Jobe JB, Smith DM, Ball K, et al. ACTIVE: a cognitive intervention trial to promote independence in older adults. *Control Clin Trials*. Aug 2001;22(4):453-479.

- 22. Ball K, Berch DB, Helmers KF, et al. Effects of cognitive training interventions with older adults: a randomized controlled trial. *JAMA*. Nov 13 2002;288(18):2271-2281.
- 23. Edwards JD, Wadley VG, Vance DE, Wood K, Roenker DL, Ball KK. The impact of speed of processing training on cognitive and everyday performance. *Aging & mental health.* May 2005;9(3):262-271.
- 24. Willis SL, Tennstedt SL, Marsiske M, et al. Long-term effects of cognitive training on everyday functional outcomes in older adults. *JAMA*. Dec 20 2006;296(23):2805-2814.
- 25. Edwards JD, Ross LA, Ackerman ML, et al. Longitudinal predictors of driving cessation among older adults from the ACTIVE clinical trial. *The journals of gerontology. Series B, Psychological sciences and social sciences.* Jan 2008;63(1):P6-12.
- 26. Edwards JD, Myers C, Ross LA, et al. The longitudinal impact of cognitive speed of processing training on driving mobility. *The Gerontologist.* Aug 2009;49(4):485-494.
- 27. Wolinsky FD, Vander Weg MW, Martin R, et al. The effect of speed-of-processing training on depressive symptoms in ACTIVE. *The journals of gerontology. Series A, Biological sciences and medical sciences.* Apr 2009;64(4):468-472.
- 28. Ball K, Edwards JD, Ross LA, McGwin G, Jr. Cognitive training decreases motor vehicle collision involvement of older drivers. *J Am Geriatr Soc.* Nov 2010;58(11):2107-2113.
- 29. Wolinsky FD, Mahncke H, Vander Weg MW, et al. Speed of processing training protects self-rated health in older adults: enduring effects observed in the multi-site ACTIVE randomized controlled trial. *International psychogeriatrics / IPA*. May 2010;22(3):470-478.
- 30. Wolinsky FD, Vander Weg MW, Martin R, et al. Does cognitive training improve internal locus of control among older adults? *The journals of gerontology. Series B, Psychological sciences and social sciences.* Sep 2010;65(5):591-598.
- 31. Belchior P, Marsiske M, Sisco SM, et al. Video game training to improve selective visual attention in older adults. *Computers in human behavior*. Jul 1 2013;29(4):1318-1324.
- 32. Jones RN, Marsiske M, Ball K, et al. The ACTIVE cognitive training interventions and trajectories of performance among older adults. *J Aging Health*. Dec 2013;25(8 Suppl):186S-208S.
- 33. Marsiske M, Dzierzewski JM, Thomas KR, et al. Race-related disparities in 5-year cognitive level and change in untrained active participants. *J Aging Health*. Dec 2013;25(8 Suppl):103S-127S.
- 34. Ross L, Edwards, JD, Ball, K. Mobility Outcomes in ACTIVE. Paper presented at: Gerontological Society of America Meetings 2013; New Orleans, LA.
- 35. Ross LA, Edwards, J. D., & Ball, K. . Mobility Outcomes in ACTIVE. Gerontological Society of America Meetings; 2013; New Orleans, LA.
- 36. Rebok GW, Ball K, Guey LT, et al. Ten-Year Effects of the Advanced Cognitive Training for Independent and Vital Elderly Cognitive Training Trial on Cognition and Everyday Functioning in Older Adults. *J Am Geriatr Soc.* Jan 13 2014.

- 37. Edwards JD, Ruva CL, O'Brien JL, Haley CB, Lister JJ. An examination of mediators of the transfer of cognitive speed of processing training to everyday functional performance. *Psychology and aging.* Jun 2013;28(2):314-321.
- 38. Edwards JD, Hauser RA, O'Connor ML, Valdes EG, Zesiewicz TA, Uc EY. Randomized trial of cognitive speed of processing training in Parkinson disease. *Neurology*. Oct 8 2013;81(15):1284-1290.
- 39. Edwards JD, Valdes EG, Peronto C, et al. The Efficacy of InSight Cognitive Training to Improve Useful Field of View Performance: A Brief Report. *The journals of gerontology. Series B, Psychological sciences and social sciences.* Nov 8 2013.
- 40. Wolinsky FD, Unverzagt FW, Smith DM, Jones R, Wright E, Tennstedt SL. The effects of the ACTIVE cognitive training trial on clinically relevant declines in health-related quality of life. *The journals of gerontology. Series B, Psychological sciences and social sciences.* Sep 2006;61(5):S281-287.
- 41. Wolinsky FD, Vander Weg MW, Howren MB, Jones MP, Dotson MM. A randomized controlled trial of cognitive training using a visual speed of processing intervention in middle aged and older adults. *PloS one*. 2013;8(5):e61624.
- 42. Singer T, Verhaeghen P, Ghisletta P, Lindenberger U, Baltes PB. The fate of cognition in very old age: six-year longitudinal findings in the Berlin Aging Study (BASE). *Psychology and aging*. Jun 2003;18(2):318-331.
- 43. Berry AS, Zanto TP, Clapp WC, et al. The influence of perceptual training on working memory in older adults. *PloS one*. 2010;5(7):e11537.
- 44. Jaeggi SM, Buschkuehl M, Jonides J, Perrig WJ. Improving fluid intelligence with training on working memory. *Proceedings of the National Academy of Sciences of the United States of America*. May 13 2008;105(19):6829-6833.
- 45. Jaeggi SM, Buschkuehl M, Perrig WJ, Meier B. The concurrent validity of the N-back task as a working memory measure. *Memory*. May 2010;18(4):394-412.
- 46. Schneider-Garces NJ, Gordon BA, Brumback-Peltz CR, et al. Span, CRUNCH, and beyond: working memory capacity and the aging brain. *Journal of cognitive neuroscience*. Apr 2010;22(4):655-669.
- 47. Brehmer Y, Rieckmann A, Bellander M, Westerberg H, Fischer H, Backman L. Neural correlates of training-related working-memory gains in old age. *Neuroimage*. Oct 15 2011;58(4):1110-1120.
- 48. Brehmer Y, Westerberg H, Backman L. Working-memory training in younger and older adults: training gains, transfer, and maintenance. *Frontiers in human neuroscience*. 2012:6:63.
- 49. Harrison PJ. The neuropathology of schizophrenia. A critical review of the data and their interpretation. *Brain.* Apr 1999;122 ( Pt 4):593-624.
- 50. Jaeggi SM, Studer-Luethi, B., Buschkuehl, M., Su, Y. F., Jonides, J., & Perrig, W. J. . The relationship between n-back performance and matrix reasoning—Implications for training and transfer. *Intelligence*. 2010;38(6):625-635.
- 51. Jaeggi SM, Buschkuehl, M., Jonides, J., & Shah, P. Cogmed and working memory training—Current challenges and the search for underlying mechanisms. *J Appl Res Mem Cogn.* 2012;1(3):211-213.

- 52. Klingberg T. Training Working Memory. *The ADHD Report: Special Issue— Focus on Assessment.* 2006;14(1):6-8.
- 53. Coull JT, Nobre AC, Frith CD. The noradrenergic alpha2 agonist clonidine modulates behavioural and neuroanatomical correlates of human attentional orienting and alerting. *Cerebral cortex*. Jan 2001;11(1):73-84.
- 54. Heilman KM, Schwartz HD, Watson RT. Hypoarousal in patients with the neglect syndrome and emotional indifference. *Neurology*. Mar 1978;28(3):229-232.
- 55. Hjaltason H, Tegner R, Tham K, Levander M, Ericson K. Sustained attention and awareness of disability in chronic neglect. *Neuropsychologia*. Dec 1996;34(12):1229-1233.
- 56. Husain M, Shapiro K, Martin J, Kennard C. Abnormal temporal dynamics of visual attention in spatial neglect patients. *Nature*. Jan 9 1997;385(6612):154-156.
- 57. Malhotra P, Coulthard EJ, Husain M. Role of right posterior parietal cortex in maintaining attention to spatial locations over time. *Brain.* Mar 2009;132(Pt 3):645-660.
- 58. Posner MI. Measuring alertness. *Annals of the New York Academy of Sciences*. 2008;1129:193-199.
- 59. Robertson IH, Mattingley JB, Rorden C, Driver J. Phasic alerting of neglect patients overcomes their spatial deficit in visual awareness. *Nature*. Sep 10 1998;395(6698):169-172.
- 60. Sturm W, Willmes K. On the functional neuroanatomy of intrinsic and phasic alertness. *Neuroimage*. Jul 2001;14(1 Pt 2):S76-84.
- 61. Thiel CM, Zilles K, Fink GR. Cerebral correlates of alerting, orienting and reorienting of visuospatial attention: an event-related fMRI study. *Neuroimage*. Jan 2004;21(1):318-328.
- 62. Thimm M, Fink GR, Kust J, Karbe H, Sturm W. Impact of alertness training on spatial neglect: a behavioural and fMRI study. *Neuropsychologia*. 2006;44(7):1230-1246.
- 63. Woods AJ, Mennemeier M, Garcia-Rill E, et al. Improvement in arousal, visual neglect, and perception of stimulus intensity following cold pressor stimulation. *Neurocase*. 2012;18(2):115-122.
- 64. Woods AJ, Philbeck JW, Chelette K, Skinner RD, Garcia-Rill E, Mennemeier M. Cold pressor stimulation diminishes P50 amplitude in normal subjects. *Acta neurobiologiae experimentalis*. 2011;71(3):348-358.
- 65. Woods AJ, Philbeck JW, Wirtz P. Hyper-arousal decreases human visual thresholds. *PloS one*. 2013;8(4):e61415.
- 66. Degutis JM, Van Vleet TM. Tonic and phasic alertness training: a novel behavioral therapy to improve spatial and non-spatial attention in patients with hemispatial neglect. *Frontiers in human neuroscience*. 2010;4.
- 67. Van Vleet TM, Hoang-duc AK, DeGutis J, Robertson LC. Modulation of non-spatial attention and the global/local processing bias. *Neuropsychologia*. Feb 2011;49(3):352-359.
- 68. Wolinsky FD, Unverzagt FW, Smith DM, Jones R, Stoddard A, Tennstedt SL. The ACTIVE cognitive training trial and health-related quality of life: protection

- that lasts for 5 years. The journals of gerontology. Series A, Biological sciences and medical sciences. Dec 2006;61(12):1324-1329.
- 69. Antal A, Fischer T, Saiote C, et al. Transcranial electrical stimulation modifies the neuronal response to psychosocial stress exposure. *Human brain mapping*. Dec 31 2013.
- 70. Arlotti M, Rahman A, Minhas P, Bikson M. Axon terminal polarization induced by weak uniform DC electric fields: a modeling study. *Conference proceedings: ...*Annual International Conference of the IEEE Engineering in Medicine and Biology Society. IEEE Engineering in Medicine and Biology Society. Conference. 2012;2012:4575-4578.
- 71. Chrysikou EG, Hamilton RH. Noninvasive brain stimulation in the treatment of aphasia: exploring interhemispheric relationships and their implications for neurorehabilitation. *Restorative neurology and neuroscience*. 2011;29(6):375-394.
- 72. Clark VP, Coffman BA, Mayer AR, et al. TDCS guided using fMRI significantly accelerates learning to identify concealed objects. *Neuroimage*. Jan 2 2012;59(1):117-128.
- 73. da Silva MC, Conti CL, Klauss J, et al. Behavioral effects of transcranial Direct Current Stimulation (tDCS) induced dorsolateral prefrontal cortex plasticity in alcohol dependence. *Journal of physiology, Paris.* Dec 2013;107(6):493-502.
- 74. Moreno-Duarte I, Morse LR, Alam M, Bikson M, Zafonte R, Fregni F. Targeted therapies using electrical and magnetic neural stimulation for the treatment of chronic pain in spinal cord injury. *Neuroimage*. Jan 15 2014;85 Pt 3:1003-1013.
- 75. Nawani H, Kalmady SV, Bose A, et al. Neural Basis of tDCS Effects on Auditory Verbal Hallucinations in Schizophrenia: A Case Report Evidence for Cortical Neuroplasticity Modulation. *The journal of ECT.* Mar 2014;30(1):e2-4.
- 76. Nitsche MA, Niehaus L, Hoffmann KT, et al. MRI study of human brain exposed to weak direct current stimulation of the frontal cortex. *Clinical neurophysiology : official journal of the International Federation of Clinical Neurophysiology.* Oct 2004;115(10):2419-2423.
- 77. Nord CL, Lally N, Charpentier CJ. Harnessing electric potential: DLPFC tDCS induces widespread brain perfusion changes. *Frontiers in systems neuroscience*. 2013;7:99.
- 78. Okano AH, Fontes EB, Montenegro RA, et al. Brain stimulation modulates the autonomic nervous system, rating of perceived exertion and performance during maximal exercise. *British journal of sports medicine*. Feb 27 2013.
- 79. Radman T, Datta A, Ramos RL, Brumberg JC, Bikson M. One-dimensional representation of a neuron in a uniform electric field. *Conference proceedings : ... Annual International Conference of the IEEE Engineering in Medicine and Biology Society. IEEE Engineering in Medicine and Biology Society. Conference.* 2009;2009:6481-6484.
- 80. Rahman A, Reato D, Arlotti M, et al. Cellular effects of acute direct current stimulation: somatic and synaptic terminal effects. *The Journal of physiology*. May 15 2013;591(Pt 10):2563-2578.
- 81. Reato D, Rahman A, Bikson M, Parra LC. Effects of weak transcranial alternating current stimulation on brain activity-a review of known mechanisms from animal studies. *Frontiers in human neuroscience*. 2013;7:687.
- 82. Sehm B, Schafer A, Kipping J, et al. Dynamic modulation of intrinsic functional connectivity by transcranial direct current stimulation. *Journal of neurophysiology*. Dec 2012;108(12):3253-3263.
- 83. Shah PP, Szaflarski JP, Allendorfer J, Hamilton RH. Induction of neuroplasticity and recovery in post-stroke aphasia by non-invasive brain stimulation. *Frontiers in human neuroscience*. 2013;7:888.
- 84. Stagg CJ, Bachtiar V, Johansen-Berg H. The role of GABA in human motor learning. *Current biology: CB.* Mar 22 2011;21(6):480-484.
- 85. Stagg CJ, Lin RL, Mezue M, et al. Widespread modulation of cerebral perfusion induced during and after transcranial direct current stimulation applied to the left dorsolateral prefrontal cortex. *J Neurosci.* Jul 10 2013;33(28):11425-11431.
- 86. Stagg CJ, Nitsche MA. Physiological basis of transcranial direct current stimulation. *The Neuroscientist: a review journal bringing neurobiology, neurology and psychiatry.* Feb 2011;17(1):37-53.
- 87. Turkeltaub PE, Benson J, Hamilton RH, Datta A, Bikson M, Coslett HB. Left lateralizing transcranial direct current stimulation improves reading efficiency. *Brain stimulation*. Jul 2012;5(3):201-207.
- 88. Woods AJ, Hamilton RH, Kranjec A, et al. Space, Time, and Causality in the Human Brain. *Neuroimage*. Feb 18 2014.
- 89. Zheng X, Alsop DC, Schlaug G. Effects of transcranial direct current stimulation (tDCS) on human regional cerebral blood flow. *Neuroimage*. Sep 1 2011;58(1):26-33.
- 90. Fregni F, Boggio PS, Santos MC, et al. Noninvasive cortical stimulation with transcranial direct current stimulation in Parkinson's disease. *Movement disorders : official journal of the Movement Disorder Society.* Oct 2006;21(10):1693-1702.
- 91. Kessler SK, Minhas P, Woods AJ, Rosen A, Gorman C, Bikson M. Dosage considerations for transcranial direct current stimulation in children: a computational modeling study. *PloS one*. 2013;8(9):e76112.
- 92. Lang N, Nitsche MA, Paulus W, Rothwell JC, Lemon RN. Effects of transcranial direct current stimulation over the human motor cortex on corticospinal and transcallosal excitability. *Experimental brain research*. Jun 2004;156(4):439-443.
- 93. Lang N, Siebner HR, Ward NS, et al. How does transcranial DC stimulation of the primary motor cortex alter regional neuronal activity in the human brain? *The European journal of neuroscience*. Jul 2005;22(2):495-504.
- 94. Liebetanz D, Nitsche MA, Tergau F, Paulus W. Pharmacological approach to the mechanisms of transcranial DC-stimulation-induced after-effects of human motor cortex excitability. *Brain.* Oct 2002;125(Pt 10):2238-2247.
- 95. Minhas P, Bikson M, Woods AJ, Rosen AR, Kessler SK. Transcranial direct current stimulation in pediatric brain: a computational modeling study. Conference proceedings: ... Annual International Conference of the IEEE Engineering in Medicine and Biology Society. IEEE Engineering in Medicine and Biology Society. Conference. 2012;2012:859-862.

- 96. Feng WW, Bowden MG, Kautz S. Review of transcranial direct current stimulation in poststroke recovery. *Topics in stroke rehabilitation*. Jan-Feb 2013;20(1):68-77.
- 97. Polanowska K, Seniow J. [Influence of transcranial direct current stimulation on cognitive functioning of patients with brain injury]. *Neurologia i neurochirurgia polska*. Nov-Dec 2010;44(6):580-590.
- 98. Schlaug G, Renga V. Transcranial direct current stimulation: a noninvasive tool to facilitate stroke recovery. *Expert review of medical devices*. Nov 2008;5(6):759-768.
- 99. Schlaug G, Renga V, Nair D. Transcranial direct current stimulation in stroke recovery. *Archives of neurology*. Dec 2008;65(12):1571-1576.
- 100. Berryhill ME, Jones KT. tDCS selectively improves working memory in older adults with more education. *Neuroscience letters*. Jul 19 2012;521(2):148-151.
- Cerruti C, Schlaug G. Anodal transcranial direct current stimulation of the prefrontal cortex enhances complex verbal associative thought. *Journal of* cognitive neuroscience. Oct 2009;21(10):1980-1987.
- 102. Dell'Osso B, Zanoni S, Ferrucci R, et al. Transcranial direct current stimulation for the outpatient treatment of poor-responder depressed patients. *European psychiatry : the journal of the Association of European Psychiatrists*. Oct 2012;27(7):513-517.
- 103. Javadi AH, Walsh V. Transcranial direct current stimulation (tDCS) of the left dorsolateral prefrontal cortex modulates declarative memory. *Brain stimulation*. Jul 2012;5(3):231-241.
- 104. Brunoni AR, Nitsche MA, Bolognini N, et al. Clinical research with transcranial direct current stimulation (tDCS): challenges and future directions. *Brain stimulation*. Jul 2012;5(3):175-195.
- 105. Cohen Kadosh R, Soskic S, Iuculano T, Kanai R, Walsh V. Modulating neuronal activity produces specific and long-lasting changes in numerical competence. *Current biology : CB.* Nov 23 2010;20(22):2016-2020.
- 106. Dockery CA, Hueckel-Weng R, Birbaumer N, Plewnia C. Enhancement of planning ability by transcranial direct current stimulation. *J Neurosci.* Jun 3 2009;29(22):7271-7277.
- 107. Hamilton RH, Chrysikou EG, Coslett B. Mechanisms of aphasia recovery after stroke and the role of noninvasive brain stimulation. *Brain and language*. Jul 2011;118(1-2):40-50.
- 108. Park SH, Seo JH, Kim YH, Ko MH. Long-term effects of transcranial direct current stimulation combined with computer-assisted cognitive training in healthy older adults. *Neuroreport*. Jan 22 2014;25(2):122-126.
- 109. Ditye T, Jacobson L, Walsh V, Lavidor M. Modulating behavioral inhibition by tDCS combined with cognitive training. *Experimental brain research*. Jun 2012;219(3):363-368.
- 110. Lesniak M, Polanowska K, Seniow J, Czlonkowska A. Effects of Repeated Anodal tDCS Coupled With Cognitive Training for Patients With Severe Traumatic Brain Injury: A Pilot Randomized Controlled Trial. The Journal of head trauma rehabilitation. Jun 10 2013.

- 111. Li SC, Schmiedek F, Huxhold O, Rocke C, Smith J, Lindenberger U. Working memory plasticity in old age: practice gain, transfer, and maintenance. *Psychology and aging*. Dec 2008;23(4):731-742.
- 112. Martin DM, Liu R, Alonzo A, et al. Can transcranial direct current stimulation enhance outcomes from cognitive training? A randomized controlled trial in healthy participants. The international journal of neuropsychopharmacology / official scientific journal of the Collegium Internationale

  Neuropsychopharmacologicum. Oct 2013;16(9):1927-1936.
- 113. Kim GW, Ko MH. Facilitation of corticospinal tract excitability by transcranial direct current stimulation combined with voluntary grip exercise. *Neuroscience letters*. Aug 26 2013;548:181-184.
- 114. Krause B, Marquez-Ruiz J, Kadosh RC. The effect of transcranial direct current stimulation: a role for cortical excitation/inhibition balance? *Frontiers in human neuroscience*. 2013;7:602.
- 115. Nitsche MA, Liebetanz D, Schlitterlau A, et al. GABAergic modulation of DC stimulation-induced motor cortex excitability shifts in humans. *The European journal of neuroscience*. May 2004;19(10):2720-2726.
- 116. Ranieri F, Podda MV, Riccardi E, et al. Modulation of LTP at rat hippocampal CA3-CA1 synapses by direct current stimulation. *Journal of neurophysiology*. Apr 2012;107(7):1868-1880.
- 117. Tremblay S, Beaule V, Lepage JF, Theoret H. Anodal transcranial direct current stimulation modulates GABAB-related intracortical inhibition in the M1 of healthy individuals. *Neuroreport*. Jan 9 2013;24(1):46-50.
- 118. Stopa EG, Butala P, Salloway S, et al. Cerebral cortical arteriolar angiopathy, vascular beta-amyloid, smooth muscle actin, Braak stage, and APOE genotype. *Stroke; a journal of cerebral circulation.* Mar 2008;39(3):814-821.
- 119. Rapp MA, Schnaider-Beeri M, Purohit DP, Perl DP, Haroutunian V, Sano M. Increased neurofibrillary tangles in patients with Alzheimer disease with comorbid depression. *Am J Geriatr Psychiatry*. Feb 2008;16(2):168-174.
- 120. Mortimer JA, Gosche KM, Riley KP, Markesbery WR, Snowdon DA. Delayed recall, hippocampal volume and Alzheimer neuropathology: findings from the Nun Study. *Neurology*. Feb 10 2004;62(3):428-432.
- 121. Braak E, Griffing K, Arai K, Bohl J, Bratzke H, Braak H. Neuropathology of Alzheimer's disease: what is new since A. Alzheimer? *Eur Arch Psychiatry Clin Neurosci.* 1999;249 Suppl 3:14-22.
- 122. Thal DR, Arendt T, Waldmann G, et al. Progression of neurofibrillary changes and PHF-tau in end-stage Alzheimer's disease is different from plaque and cortical microglial pathology. *Neurobiol Aging*. Nov-Dec 1998;19(6):517-525.
- 123. Thal DR, Hartig W, Schober R. Stage-correlated distribution of type 1 and 2 dystrophic neurites in cortical and hippocampal plaques in Alzheimer's disease. *J Hirnforsch.* 1998;39(2):175-181.
- 124. Mizukami K, Grayson DR, Ikonomovic MD, Sheffield R, Armstrong DM. GABAA receptor beta 2 and beta 3 subunits mRNA in the hippocampal formation of aged human brain with Alzheimer-related neuropathology. *Brain Res Mol Brain Res.* May 1998;56(1-2):268-272.

- 125. Jellinger KA, Bancher C. Senile dementia with tangles (tangle predominant form of senile dementia). *Brain Pathol.* Apr 1998;8(2):367-376.
- 126. Nagy Z, Vatter-Bittner B, Braak H, et al. Staging of Alzheimer-type pathology: an interrater-intrarater study. *Dement Geriatr Cogn Disord*. Jul-Aug 1997;8(4):248-251.
- 127. Braak H, Braak E. Evolution of the neuropathology of Alzheimer's disease. *Acta Neurol Scand Suppl.* 1996;165:3-12.
- 128. Knopman DS, Parisi JE, Salviati A, et al. Neuropathology of cognitively normal elderly. *J Neuropathol Exp Neurol*. Nov 2003;62(11):1087-1095.
- 129. Raz N, Schmiedek F, Rodrigue KM, Kennedy KM, Lindenberger U, Lovden M. Differential brain shrinkage over 6 months shows limited association with cognitive practice. *Brain Cogn.* Jul 2013;82(2):171-180.
- 130. Fjell AM, Westlye LT, Grydeland H, et al. Critical ages in the life course of the adult brain: nonlinear subcortical aging. *Neurobiol Aging*. Oct 2013;34(10):2239-2247
- 131. Raz N, Yang YQ, Rodrigue KM, Kennedy KM, Lindenberger U, Ghisletta P. White matter deterioration in 15 months: latent growth curve models in healthy adults. *Neurobiol Aging*. Feb 2012;33(2):429 e421-425.
- 132. Rodrigue KM, Haacke EM, Raz N. Differential effects of age and history of hypertension on regional brain volumes and iron. *Neuroimage*. Jan 15 2011;54(2):750-759.
- 133. Raz N, Ghisletta P, Rodrigue KM, Kennedy KM, Lindenberger U. Trajectories of brain aging in middle-aged and older adults: regional and individual differences. *Neuroimage*. Jun 2010;51(2):501-511.
- 134. Burgmans S, van Boxtel MP, Gronenschild EH, et al. Multiple indicators of agerelated differences in cerebral white matter and the modifying effects of hypertension. *Neuroimage*. Feb 1 2010;49(3):2083-2093.
- 135. Kennedy KM, Rodrigue KM, Head D, Gunning-Dixon F, Raz N. Neuroanatomical and cognitive mediators of age-related differences in perceptual priming and learning. *Neuropsychology*. Jul 2009;23(4):475-491.
- 136. Head D, Rodrigue KM, Kennedy KM, Raz N. Neuroanatomical and cognitive mediators of age-related differences in episodic memory. *Neuropsychology*. Jul 2008;22(4):491-507.
- 137. Kennedy KM, Erickson KI, Rodrigue KM, et al. Age-related differences in regional brain volumes: a comparison of optimized voxel-based morphometry to manual volumetry. *Neurobiol Aging*. Oct 2009;30(10):1657-1676.
- 138. Raz N, Rodrigue KM, Haacke EM. Brain aging and its modifiers: insights from in vivo neuromorphometry and susceptibility weighted imaging. *Annals of the New York Academy of Sciences*. Feb 2007;1097:84-93.
- 139. Erickson KI, Colcombe SJ, Raz N, et al. Selective sparing of brain tissue in postmenopausal women receiving hormone replacement therapy. *Neurobiol Aging*. Aug-Sep 2005;26(8):1205-1213.
- 140. Raz N, Lindenberger U, Rodrigue KM, et al. Regional brain changes in aging healthy adults: general trends, individual differences and modifiers. *Cerebral cortex*. Nov 2005;15(11):1676-1689.

- 141. Raz N, Gunning-Dixon FM, Head D, Dupuis JH, Acker JD. Neuroanatomical correlates of cognitive aging: evidence from structural magnetic resonance imaging. *Neuropsychology*. Jan 1998;12(1):95-114.
- 142. Raz N, Gunning FM, Head D, et al. Selective aging of the human cerebral cortex observed in vivo: differential vulnerability of the prefrontal gray matter. *Cerebral cortex*. Apr-May 1997;7(3):268-282.
- 143. Raz N, Torres IJ, Acker JD. Age, gender, and hemispheric differences in human striatum: a quantitative review and new data from in vivo MRI morphometry. *Neurobiol Learn Mem.* Mar 1995;63(2):133-142.
- 144. Raz N, Torres IJ, Briggs SD, et al. Selective neuroanatomic abnormalities in Down's syndrome and their cognitive correlates: evidence from MRI morphometry. *Neurology*. Feb 1995;45(2):356-366.
- 145. Brickman AM, Provenzano FA, Muraskin J, et al. Regional white matter hyperintensity volume, not hippocampal atrophy, predicts incident Alzheimer disease in the community. *Archives of neurology*. Dec 2012;69(12):1621-1627.
- 146. Zimmerman ME, Brickman AM, Paul RH, et al. The relationship between frontal gray matter volume and cognition varies across the healthy adult lifespan. *Am J Geriatr Psychiatry*. Oct 2006;14(10):823-833.
- 147. Brickman AM, Habeck C, Zarahn E, Flynn J, Stern Y. Structural MRI covariance patterns associated with normal aging and neuropsychological functioning. *Neurobiol Aging.* Feb 2007;28(2):284-295.
- 148. Paul RH, Haque O, Gunstad J, et al. Subcortical hyperintensities impact cognitive function among a select subset of healthy elderly. *Arch Clin Neuropsychol.* Aug 2005;20(6):697-704.
- 149. Tate DF, Jefferson AL, Brickman AM, et al. Regional White Matter Signal Abnormalities and Cognitive Correlates Among Geriatric Patients with Treated Cardiovascular Disease. *Brain Imaging Behav.* Sep 1 2008;2(3):200-206.
- 150. Jefferson AL, Tate DF, Poppas A, et al. Lower cardiac output is associated with greater white matter hyperintensities in older adults with cardiovascular disease. *J Am Geriatr Soc.* Jul 2007;55(7):1044-1048.
- 151. Miller LA, Gunstad J, Spitznagel MB, et al. CAMTA1 T polymorphism is associated with neuropsychological test performance in older adults with cardiovascular disease. *Psychogeriatrics*. Sep 2011;11(3):135-140.
- 152. Cohen RA, Poppas A, Forman DE, et al. Vascular and cognitive functions associated with cardiovascular disease in the elderly. *J Clin Exp Neuropsychol.* Jan 2009;31(1):96-110.
- 153. Haley AP, Sweet LH, Gunstad J, et al. Verbal working memory and atherosclerosis in patients with cardiovascular disease: an fMRI study. *J Neuroimaging*. Jul 2007;17(3):227-233.
- 154. Hoth KF, Tate DF, Poppas A, et al. Endothelial function and white matter hyperintensities in older adults with cardiovascular disease. *Stroke; a journal of cerebral circulation*. Feb 2007;38(2):308-312.
- 155. Garrett KD, Browndyke JN, Whelihan W, et al. The neuropsychological profile of vascular cognitive impairment--no dementia: comparisons to patients at risk for cerebrovascular disease and vascular dementia. *Arch Clin Neuropsychol.* Sep 2004;19(6):745-757.

- 156. Alosco ML, Gunstad J, Jerskey BA, et al. The adverse effects of reduced cerebral perfusion on cognition and brain structure in older adults with cardiovascular disease. *Brain Behav.* Nov 2013;3(6):626-636.
- 157. Irani F, Sweet LH, Haley AP, et al. A fMRI Study of Verbal Working Memory, Cardiac Output, and Ejection Fraction in Elderly Patients with Cardiovascular Disease. *Brain Imaging Behav.* Dec 2009;3(4):350-357.
- 158. Haley AP, Hoth KF, Gunstad J, et al. Subjective cognitive complaints relate to white matter hyperintensities and future cognitive decline in patients with cardiovascular disease. *Am J Geriatr Psychiatry*. Nov 2009;17(11):976-985.
- 159. Gunstad J, Bausserman L, Paul RH, et al. C-reactive protein, but not homocysteine, is related to cognitive dysfunction in older adults with cardiovascular disease. *J Clin Neurosci.* Jun 2006;13(5):540-546.
- 160. Gunstad J, Cohen RA, Tate DF, et al. Blood pressure variability and white matter hyperintensities in older adults with cardiovascular disease. *Blood Press*. 2005;14(6):353-358.
- 161. Raz N, Williamson A, Gunning-Dixon F, Head D, Acker JD. Neuroanatomical and cognitive correlates of adult age differences in acquisition of a perceptual-motor skill. *Microsc Res Tech.* Oct 1 2000;51(1):85-93.
- 162. Brickman AM, Zimmerman ME, Paul RH, et al. Regional white matter and neuropsychological functioning across the adult lifespan. *Biol Psychiatry*. Sep 1 2006;60(5):444-453.
- 163. Brickman AM. Contemplating Alzheimer's disease and the contribution of white matter hyperintensities. *Curr Neurol Neurosci Rep.* Dec 2013;13(12):415.
- 164. Brickman AM, Buchsbaum MS, Shihabuddin L, Hazlett EA, Borod JC, Mohs RC. Striatal size, glucose metabolic rate, and verbal learning in normal aging. *Brain Res Cogn Brain Res*. Jun 2003;17(1):106-116.
- 165. Brickman AM, Paul RH, Cohen RA, et al. Category and letter verbal fluency across the adult lifespan: relationship to EEG theta power. *Arch Clin Neuropsychol.* Jul 2005;20(5):561-573.
- 166. Brickman AM, Schupf N, Manly JJ, et al. Brain morphology in older African Americans, Caribbean Hispanics, and whites from northern Manhattan. *Archives of neurology*. Aug 2008;65(8):1053-1061.
- 167. Brickman AM, Sneed JR, Provenzano FA, et al. Quantitative approaches for assessment of white matter hyperintensities in elderly populations. *Psychiatry Res.* Aug 30 2011;193(2):101-106.
- 168. Cohen R, Sweet LH. *Neuroimaging in Behavioral Medicine and Clinical Neuroscience*. New York, NY: Springer Publishing; 2012.
- 169. Clark US, Cohen RA, Sweet LH, et al. Effects of HIV and early life stress on amygdala morphometry and neurocognitive function. *J Int Neuropsychol Soc.* Jul 2012;18(4):657-668.
- 170. Sweet LH, Hassenstab JJ, McCaffery JM, et al. Brain response to food stimulation in obese, normal weight, and successful weight loss maintainers. *Obesity (Silver Spring)*. Nov 2012;20(11):2220-2225.
- 171. Sweet LH, Mulligan RC, Finnerty CE, et al. Effects of nicotine withdrawal on verbal working memory and associated brain response. *Psychiatry Res.* Jul 30 2010;183(1):69-74.

- 172. McCaffery JM, Haley AP, Sweet LH, et al. Differential functional magnetic resonance imaging response to food pictures in successful weight-loss maintainers relative to normal-weight and obese controls. *Am J Clin Nutr.* Oct 2009;90(4):928-934.
- 173. Browndyke JN, Paskavitz J, Sweet LH, et al. Neuroanatomical correlates of malingered memory impairment: event-related fMRI of deception on a recognition memory task. *Brain Inj.* Jun 2008;22(6):481-489.
- 174. David SP, Munafo MR, Johansen-Berg H, et al. Effects of Acute Nicotine Abstinence on Cue-elicited Ventral Striatum/Nucleus Accumbens Activation in Female Cigarette Smokers: A Functional Magnetic Resonance Imaging Study. *Brain Imaging Behav.* Dec 2007;1(3-4):43-57.
- 175. Sweet LH, Paskavitz JF, Haley AP, et al. Imaging phonological similarity effects on verbal working memory. *Neuropsychologia*. Mar 7 2008;46(4):1114-1123.
- 176. Sweet LH, Paskavitz JF, O'Connor MJ, Browndyke JN, Wellen JW, Cohen RA. FMRI correlates of the WAIS-III symbol search subtest. *J Int Neuropsychol Soc.* Jul 2005;11(4):471-476.
- 177. Sweet LH, Rao SM, Primeau M, Durgerian S, Cohen RA. Functional magnetic resonance imaging response to increased verbal working memory demands among patients with multiple sclerosis. *Human brain mapping*. Jan 2006;27(1):28-36.
- 178. Sweet LH, Rao SM, Primeau M, Mayer AR, Cohen RA. Functional magnetic resonance imaging of working memory among multiple sclerosis patients. *J Neuroimaging*. Apr 2004;14(2):150-157.
- 179. Sweet LH, Paul RH, Cohen RA, et al. Neuroimaging correlates of dementia rating scale performance at baseline and 12-month follow-up among patients with vascular dementia. *J Geriatr Psychiatry Neurol*. Dec 2003;16(4):240-244.
- 180. Davis SW, Kragel JE, Madden DJ, Cabeza R. The architecture of cross-hemispheric communication in the aging brain: linking behavior to functional and structural connectivity. *Cerebral cortex*. Jan 2012;22(1):232-242.
- 181. Madden DJ, Costello MC, Dennis NA, et al. Adult age differences in functional connectivity during executive control. *Neuroimage*. Aug 15 2010;52(2):643-657.
- 182. Davis SW, Dennis NA, Buchler NG, White LE, Madden DJ, Cabeza R. Assessing the effects of age on long white matter tracts using diffusion tensor tractography. *Neuroimage.* Jun 2009;46(2):530-541.
- 183. Davis SW, Dennis NA, Daselaar SM, Fleck MS, Cabeza R. Que PASA? The posterior-anterior shift in aging. *Cerebral cortex*. May 2008;18(5):1201-1209.
- 184. Chang L, Holt JL, Yakupov R, Jiang CS, Ernst T. Lower cognitive reserve in the aging human immunodeficiency virus-infected brain. *Neurobiol Aging*. Apr 2013;34(4):1240-1253.
- 185. Chang L, Lee P, Yiannoutsos C, et al. A multicenter In Vivo Proton MRS study of HIV-associated brain injury and the effects of aging. HIV MRS Consortium; Submitted.
- 186. Chang L, Speck O, Miller EN, et al. Neural correlates of attention and working memory deficits in HIV patients. *Neurology*. Sep 25 2001;57(6):1001-1007.

- 187. Chang L, Wong V, Nakama H, et al. Greater than age-related changes in brain diffusion of HIV patients after 1 year. *J Neuroimmune Pharmacol*. Dec 2008;3(4):265-274.
- 188. Ernst T, Chang L, Jovicich J, Ames N, Arnold S. Abnormal brain activation on functional MRI in cognitively asymptomatic HIV patients. *Neurology*. Nov 12 2002;59(9):1343-1349.
- 189. Ernst T, Itti E, Itti L, Chang L. Changes in cerebral metabolism are detected prior to perfusion changes in early HIV-CMC: A coregistered (1)H MRS and SPECT study. *J Magn Reson Imaging*. Dec 2000;12(6):859-865.
- 190. Ernst T, Yakupov R, Nakama H, et al. Declined neural efficiency in cognitively stable human immunodeficiency virus patients. *Ann Neurol.* Mar 2009;65(3):316-325.
- 191. Watanabe T, Shiino A, Akiguchi I. Absolute quantification in proton magnetic resonance spectroscopy is useful to differentiate amnesic mild cognitive impairment from Alzheimer's disease and healthy aging. *Dement Geriatr Cogn Disord*. 2010;30(1):71-77.
- 192. Ding B, Chen KM, Ling HW, et al. Diffusion tensor imaging correlates with proton magnetic resonance spectroscopy in posterior cingulate region of patients with Alzheimer's disease. *Dement Geriatr Cogn Disord*. 2008;25(3):218-225.
- Metastasio A, Rinaldi P, Tarducci R, et al. Conversion of MCI to dementia: Role of proton magnetic resonance spectroscopy. *Neurobiol Aging*. Jul 2006;27(7):926-932.
- 194. Ackl N, Ising M, Schreiber YA, Atiya M, Sonntag A, Auer DP. Hippocampal metabolic abnormalities in mild cognitive impairment and Alzheimer's disease. *Neuroscience letters*. Aug 12-19 2005;384(1-2):23-28.
- 195. Modrego PJ, Fayed N, Pina MA. Conversion from mild cognitive impairment to probable Alzheimer's disease predicted by brain magnetic resonance spectroscopy. *Am J Psychiatry*. Apr 2005;162(4):667-675.
- 196. Frederick BD, Lyoo IK, Satlin A, et al. In vivo proton magnetic resonance spectroscopy of the temporal lobe in Alzheimer's disease. *Prog Neuropsychopharmacol Biol Psychiatry.* Dec 2004;28(8):1313-1322.
- 197. Pilatus U, Lais C, Rochmont Adu M, et al. Conversion to dementia in mild cognitive impairment is associated with decline of N-actylaspartate and creatine as revealed by magnetic resonance spectroscopy. *Psychiatry Res.* Jul 15 2009;173(1):1-7.
- 198. Waldman AD, Rai GS. The relationship between cognitive impairment and in vivo metabolite ratios in patients with clinical Alzheimer's disease and vascular dementia: a proton magnetic resonance spectroscopy study. *Neuroradiology*. Aug 2003;45(8):507-512.
- 199. Pagonabarraga J, Gomez-Anson B, Rotger R, et al. Spectroscopic changes associated with mild cognitive impairment and dementia in Parkinson's disease. *Dement Geriatr Cogn Disord*. 2012;34(5-6):312-318.
- 200. Gasparovic C, Prestopnik J, Thompson J, et al. 1H-MR spectroscopy metabolite levels correlate with executive function in vascular cognitive impairment. *J Neurol Neurosurg Psychiatry*. Jul 2013;84(7):715-721.

- 201. Wang S, Yuan J, Guo X, et al. Neurochemical correlates of cognitive dysfunction in patients with leukoaraiosis: a proton magnetic resonance spectroscopy study. *Neurol Res.* Dec 2012;34(10):989-997.
- 202. Griffith HR, Stewart CC, den Hollander JA. Proton magnetic resonance spectroscopy in dementias and mild cognitive impairment. *Int Rev Neurobiol.* 2009;84:105-131.
- 203. Ross AJ, Sachdev PS, Wen W, Valenzuela MJ, Brodaty H. 1H MRS in stroke patients with and without cognitive impairment. *Neurobiol Aging*. Jun 2005;26(6):873-882.
- 204. Chang L, Lee PL, Yiannoutsos CT, et al. A multicenter in vivo proton-MRS study of HIV-associated dementia and its relationship to age. *Neuroimage*. Dec 2004;23(4):1336-1347.
- Lee PL, Yiannoutsos CT, Ernst T, et al. A multi-center 1H MRS study of the AIDS dementia complex: validation and preliminary analysis. *J Magn Reson Imaging*. Jun 2003;17(6):625-633.
- 206. Yiannoutsos CT, Ernst T, Chang L, et al. Regional patterns of brain metabolites in AIDS dementia complex. *Neuroimage*. Nov 2004;23(3):928-935.
- 207. Hua X, Boyle CP, Harezlak J, et al. Disrupted cerebral metabolite levels and lower nadir CD4 + counts are linked to brain volume deficits in 210 HIV-infected patients on stable treatment. *Neuroimage Clin.* 2013;3:132-142.
- 208. Harezlak J, Buchthal S, Taylor M, et al. Persistence of HIV-associated cognitive impairment, inflammation, and neuronal injury in era of highly active antiretroviral treatment. *AIDS*. Mar 13 2011;25(5):625-633.
- 209. Cohen RA, Harezlak J, Gongvatana A, et al. Cerebral metabolite abnormalities in human immunodeficiency virus are associated with cortical and subcortical volumes. *Journal of neurovirology.* Nov 2010;16(6):435-444.
- 210. Paul RH, Ernst T, Brickman AM, et al. Relative sensitivity of magnetic resonance spectroscopy and quantitative magnetic resonance imaging to cognitive function among nondemented individuals infected with HIV. *J Int Neuropsychol Soc.* Sep 2008;14(5):725-733.
- 211. Paul RH, Gunstad J, Cooper N, et al. Cross-cultural assessment of neuropsychological performance and electrical brain function measures: additional validation of an international brain database. *Int J Neurosci.* Apr 2007;117(4):549-568.
- 212. Watanabe M, Maemura K, Kanbara K, Tamayama T, Hayasaki H. GABA and GABA receptors in the central nervous system and other organs. *Int Rev Cytol.* 2002;213:1-47.
- 213. Szabadics J, Varga C, Molnar G, Olah S, Barzo P, Tamas G. Excitatory effect of GABAergic axo-axonic cells in cortical microcircuits. *Science*. Jan 13 2006;311(5758):233-235.
- 214. Foster TC, Sharrow KM, Kumar A, Masse J. Interaction of age and chronic estradiol replacement on memory and markers of brain aging. *Neurobiol Aging*. Oct 2003;24(6):839-852.
- 215. Foster TC, Kumar A. Calcium dysregulation in the aging brain. *The Neuroscientist: a review journal bringing neurobiology, neurology and psychiatry.* Aug 2002;8(4):297-301.

- 216. Foster TC, Sharrow KM, Masse JR, Norris CM, Kumar A. Calcineurin links Ca2+ dysregulation with brain aging. *J Neurosci.* Jun 1 2001;21(11):4066-4073.
- 217. Foster TC. Involvement of hippocampal synaptic plasticity in age-related memory decline. *Brain Res Brain Res Rev.* Nov 1999;30(3):236-249.
- 218. Foster TC, Norris CM. Age-associated changes in Ca(2+)-dependent processes: relation to hippocampal synaptic plasticity. *Hippocampus*. 1997;7(6):602-612.
- Baumgartner BJ, Harvey RJ, Darlison MG, Barnes EM, Jr. Developmental upregulation and agonist-dependent down-regulation of GABAA receptor subunit mRNAs in chick cortical neurons. *Brain Res Mol Brain Res*. Oct 1994;26(1-2):9-17.
- 220. Green EJ, Barnes CA, McNaughton BL. Behavioral state dependence of homoand hetero-synaptic modulation of dentate gyrus excitability. *Experimental brain* research. 1993;93(1):55-65.
- 221. Mizumori SJ, Barnes CA, McNaughton BL. Differential effects of age on subpopulations of hippocampal theta cells. *Neurobiol Aging*. Nov-Dec 1992;13(6):673-679.
- 222. Burke SN, Barnes CA. Senescent synapses and hippocampal circuit dynamics. *Trends Neurosci.* Mar 2010;33(3):153-161.
- 223. Burke SN, Maurer AP, Yang Z, Navratilova Z, Barnes CA. Glutamate receptor-mediated restoration of experience-dependent place field expansion plasticity in aged rats. *Behav Neurosci.* Jun 2008;122(3):535-548.
- 224. Barnes J, Hinkley L, Masters S, Boubert L. Visual memory transformations in dyslexia. *Percept Mot Skills*. Jun 2007;104(3 Pt 1):881-891.
- 225. Barnes P, Good M. Impaired Pavlovian cued fear conditioning in Tg2576 mice expressing a human mutant amyloid precursor protein gene. *Behav Brain Res.* Feb 10 2005;157(1):107-117.
- 226. Barnes DE, Tager IB, Satariano WA, Yaffe K. The relationship between literacy and cognition in well-educated elders. *The journals of gerontology. Series A, Biological sciences and medical sciences.* Apr 2004;59(4):390-395.
- 227. Barnes CA. Long-term potentiation and the ageing brain. *Philos Trans R Soc Lond B Biol Sci.* Apr 29 2003;358(1432):765-772.
- 228. Barnes CA, Rao G, Orr G. Age-related decrease in the Schaffer collateralevoked EPSP in awake, freely behaving rats. *Neural Plast.* 2000;7(3):167-178.
- 229. Barnes CA, Rao G, Houston FP. LTP induction threshold change in old rats at the perforant path--granule cell synapse. *Neurobiol Aging*. Sep-Oct 2000;21(5):613-620.
- 230. Barnes CA, Rao G, Shen J. Age-related decrease in the N-methyl-D-aspartateR-mediated excitatory postsynaptic potential in hippocampal region CA1. *Neurobiol Aging*. Jul-Aug 1997;18(4):445-452.
- 231. Rao G, Barnes CA, McNaughton BL. Effects of age on L-glutamate-induced depolarization in three hippocampal subfields. *Neurobiol Aging*. Jan-Feb 1993;14(1):27-33.
- 232. Nelson HE, Pantelis C, Carruthers K, Speller J, Baxendale S, Barnes TR. Cognitive functioning and symptomatology in chronic schizophrenia. *Psychol Med.* May 1990;20(2):357-365.

- 233. Barnes CA. Effects of aging on the dynamics of information processing and synaptic weight changes in the mammalian hippocampus. *Prog Brain Res.* 1990;86:89-104.
- 234. Barnes CA. Aging and the physiology of spatial memory. *Neurobiol Aging*. Sep-Dec 1988;9(5-6):563-568.
- 235. Barnes CA. Memory deficits associated with senescence: a neurophysiological and behavioral study in the rat. *J Comp Physiol Psychol*. Feb 1979;93(1):74-104.
- 236. Alexander GE, Ryan L, Bowers D, et al. Characterizing cognitive aging in humans with links to animal models. *Front Aging Neurosci.* 2012;4:21.
- 237. Bizon JL, Foster TC, Alexander GE, Glisky EL. Characterizing cognitive aging of working memory and executive function in animal models. *Front Aging Neurosci.* 2012;4:19.
- 238. Roberson ED, Defazio RA, Barnes CA, et al. Challenges and opportunities for characterizing cognitive aging across species. *Front Aging Neurosci.* 2012;4:6.
- 239. Nilsen LH, Melo TM, Saether O, Witter MP, Sonnewald U. Altered neurochemical profile in the McGill-R-Thy1-APP rat model of Alzheimer's disease: a longitudinal in vivo 1 H MRS study. *J Neurochem*. Nov 2012;123(4):532-541.
- 240. Martin WR. MR spectroscopy in neurodegenerative disease. *Mol Imaging Biol.* Jul-Aug 2007;9(4):196-203.
- 241. Broccardo C, Nieoullon V, Amin R, et al. ABCA2 is a marker of neural progenitors and neuronal subsets in the adult rodent brain. *J Neurochem.* Apr 2006;97(2):345-355.
- 242. Wang H, Lian K, Han B, et al. Age-Related Alterations in the Metabolic Profile in the Hippocampus of the Senescence-Accelerated Mouse Prone 8: A Spontaneous Alzheimer's Disease Mouse Model. *J Alzheimers Dis.* Nov 27 2013.
- 243. Paul SM, Doherty JJ, Robichaud AJ, et al. The major brain cholesterol metabolite 24(S)-hydroxycholesterol is a potent allosteric modulator of N-methyl-D-aspartate receptors. *J Neurosci*. Oct 30 2013;33(44):17290-17300.
- 244. Nilsen LH, Rae C, Ittner LM, Gotz J, Sonnewald U. Glutamate metabolism is impaired in transgenic mice with tau hyperphosphorylation. *J Cereb Blood Flow Metab*. May 2013;33(5):684-691.
- 245. Ferchmin PA, Perez D, Castro Alvarez W, Penzo MA, Maldonado HM, Eterovic VA. gamma-Aminobutyric acid type A receptor inhibition triggers a nicotinic neuroprotective mechanism. *J Neurosci Res.* Mar 2013;91(3):416-425.
- 246. Koh MT, Rosenzweig-Lipson S, Gallagher M. Selective GABA(A) alpha5 positive allosteric modulators improve cognitive function in aged rats with memory impairment. *Neuropharmacology*. Jan 2013;64:145-152.
- 247. Leon-Espinosa G, DeFelipe J, Munoz A. Effects of amyloid-beta plaque proximity on the axon initial segment of pyramidal cells. *J Alzheimers Dis.* 2012;29(4):841-852.
- 248. Krantic S, Isorce N, Mechawar N, et al. Hippocampal GABAergic neurons are susceptible to amyloid-beta toxicity in vitro and are decreased in number in the Alzheimer's disease TgCRND8 mouse model. *J Alzheimers Dis.* 2012;29(2):293-308.

- 249. Poil SS, Jansen R, van Aerde K, et al. Fast network oscillations in vitro exhibit a slow decay of temporal auto-correlations. *The European journal of neuroscience*. Aug 2011;34(3):394-403.
- 250. Li G, Bien-Ly N, Andrews-Zwilling Y, et al. GABAergic interneuron dysfunction impairs hippocampal neurogenesis in adult apolipoprotein E4 knockin mice. *Cell Stem Cell.* Dec 4 2009;5(6):634-645.
- 251. Rangel A, Madronal N, Gruart A, et al. Regulation of GABA(A) and glutamate receptor expression, synaptic facilitation and long-term potentiation in the hippocampus of prion mutant mice. *PloS one*. 2009;4(10):e7592.
- 252. Molinaro G, Battaglia G, Riozzi B, et al. Memantine treatment reduces the expression of the K(+)/Cl(-) cotransporter KCC2 in the hippocampus and cerebral cortex, and attenuates behavioural responses mediated by GABA(A) receptor activation in mice. *Brain Res.* Apr 10 2009;1265:75-79.
- 253. Matsuyama S, Taniguchi T, Kadoyama K, Matsumoto A. Long-term potentiation-like facilitation through GABAA receptor blockade in the mouse dentate gyrus in vivo. *Neuroreport*. Dec 3 2008;19(18):1809-1813.
- 254. Yuk DY, Lee YK, Nam SY, et al. Reduced anxiety in the mice expressing mutant (N141I) presenilin 2. *J Neurosci Res.* Feb 2009;87(2):522-531.
- 255. Albuquerque EX, Pereira EF, Mike A, Eisenberg HM, Maelicke A, Alkondon M. Neuronal nicotinic receptors in synaptic functions in humans and rats: physiological and clinical relevance. *Behav Brain Res.* Aug 2000;113(1-2):131-141.
- 256. Alkondon M, Pereira EF, Yu P, et al. Targeted deletion of the kynurenine aminotransferase ii gene reveals a critical role of endogenous kynurenic acid in the regulation of synaptic transmission via alpha7 nicotinic receptors in the hippocampus. *J Neurosci*. May 12 2004;24(19):4635-4648.
- 257. Edgar PF, Schonberger SJ, Dean B, Faull RL, Kydd R, Cooper GJ. A comparative proteome analysis of hippocampal tissue from schizophrenic and Alzheimer's disease individuals. *Mol Psychiatry*. Mar 1999;4(2):173-178.
- 258. Griguoli M, Cherubini E. Regulation of hippocampal inhibitory circuits by nicotinic acetylcholine receptors. *The Journal of physiology.* Feb 15 2012;590(Pt 4):655-666.
- 259. Uehara T, Sumiyoshi T, Hattori H, et al. T-817MA, a novel neurotrophic agent, ameliorates loss of GABAergic parvalbumin-positive neurons and sensorimotor gating deficits in rats transiently exposed to MK-801 in the neonatal period. *J Psychiatr Res.* May 2012;46(5):622-629.
- 260. Tao R, Li C, Newburn EN, et al. Transcript-specific associations of SLC12A5 (KCC2) in human prefrontal cortex with development, schizophrenia, and affective disorders. *J Neurosci.* Apr 11 2012;32(15):5216-5222.
- 261. Pattwell SS, Bath KG, Perez-Castro R, Lee FS, Chao MV, Ninan I. The BDNF Val66Met polymorphism impairs synaptic transmission and plasticity in the infralimbic medial prefrontal cortex. *J Neurosci*. Feb 15 2012;32(7):2410-2421.
- 262. Vinkers CH, Oosting RS, van Bogaert MJ, Olivier B, Groenink L. Early-life blockade of 5-HT(1A) receptors alters adult anxiety behavior and benzodiazepine sensitivity. *Biol Psychiatry*. Feb 15 2010;67(4):309-316.

- 263. Miczek KA, Yap JJ, Covington HE, 3rd. Social stress, therapeutics and drug abuse: preclinical models of escalated and depressed intake. *Pharmacol Ther.* Nov 2008;120(2):102-128.
- 264. Hoschl C, Hajek T. Hippocampal damage mediated by corticosteroids--a neuropsychiatric research challenge. *Eur Arch Psychiatry Clin Neurosci.* 2001;251 Suppl 2:II81-88.
- 265. Motohashi N, Ikawa K, Kariya T. GABAB receptors are up-regulated by chronic treatment with lithium or carbamazepine. GABA hypothesis of affective disorders? *Eur J Pharmacol.* Jul 4 1989;166(1):95-99.
- 266. Martin P, Pichat P, Massol J, Soubrie P, Lloyd KG, Puech AJ. Decreased GABA B receptors in helpless rats: reversal by tricyclic antidepressants. *Neuropsychobiology*. 1989;22(4):220-224.
- 267. Lloyd KG, Morselli PL, Bartholini G. GABA and affective disorders. *Med Biol.* 1987;65(2-3):159-165.
- 268. Long Z, Li XR, Xu J, et al. Thalamic GABA Predicts Fine Motor Performance in Manganese-Exposed Smelter Workers. *PloS one.* 2014;9(2):e88220.
- 269. Mullins PG, McGonigle DJ, O'Gorman RL, et al. Current practice in the use of MEGA-PRESS spectroscopy for the detection of GABA. *Neuroimage*. Feb 1 2014:86:43-52.
- 270. Shaw A, Brealy J, Richardson H, et al. Marked reductions in visual evoked responses but not gamma-aminobutyric acid concentrations or gamma-band measures in remitted depression. *Biol Psychiatry*. Apr 1 2013;73(7):691-698.
- 271. Foerster BR, Callaghan BC, Petrou M, Edden RA, Chenevert TL, Feldman EL. Decreased motor cortex gamma-aminobutyric acid in amyotrophic lateral sclerosis. *Neurology*. May 15 2012;78(20):1596-1600.
- 272. Stone JM, Dietrich C, Edden R, et al. Ketamine effects on brain GABA and glutamate levels with 1H-MRS: relationship to ketamine-induced psychopathology. *Mol Psychiatry*. Jul 2012;17(7):664-665.
- 273. Dydak U, Jiang YM, Long LL, et al. In vivo measurement of brain GABA concentrations by magnetic resonance spectroscopy in smelters occupationally exposed to manganese. *Environ Health Perspect.* Feb 2011;119(2):219-224.
- 274. Edden RA, Puts NA, Barker PB. Macromolecule-suppressed GABA-edited magnetic resonance spectroscopy at 3T. *Magn Reson Med.* Sep 2012;68(3):657-661.
- 275. Edden RA, Crocetti D, Zhu H, Gilbert DL, Mostofsky SH. Reduced GABA concentration in attention-deficit/hyperactivity disorder. *Arch Gen Psychiatry*. Jul 2012;69(7):750-753.
- 276. Michels L, Martin E, Klaver P, et al. Frontal GABA levels change during working memory. *PloS one.* 2012;7(4):e31933.
- 277. Edden RA, Intrapiromkul J, Zhu H, Cheng Y, Barker PB. Measuring T2 in vivo with J-difference editing: application to GABA at 3 Tesla. *J Magn Reson Imaging*. Jan 2012;35(1):229-234.
- 278. Edden RA, Barker PB. If J doesn't evolve, it won't J-resolve: J-PRESS with bandwidth-limited refocusing pulses. *Magn Reson Med.* Jun 2011;65(6):1509-1514.

- 279. Sisco SM, Marsiske M, Gross AL, Rebok GW. The influence of cognitive training on older adults' recall for short stories. *J Aging Health*. Dec 2013;25(8 Suppl):230S-248S.
- 280. Payne BR, Gross AL, Parisi JM, et al. Modelling longitudinal changes in older adults' memory for spoken discourse: Findings from the ACTIVE cohort. *Memory*. Dec 4 2013.
- 281. Merzenich M. POSIT Science. 2014; http://www.positscience.com.
- 282. Nadeau SE, Wu SS. CIMT as a behavioral engine in research on physiological adjuvants to neurorehabilitation: the challenge of merging animal and human research. *NeuroRehabilitation*. 2006;21(2):107-130.
- 283. Batsikadze G, Moliadze V, Paulus W, Kuo MF, Nitsche MA. Partially non-linear stimulation intensity-dependent effects of direct current stimulation on motor cortex excitability in humans. *The Journal of physiology.* Apr 1 2013;591(Pt 7):1987-2000.
- 284. Trahan DE, Larrabee GJ, Quintana JW. Visual recognition memory in normal adults and patients with unilateral vascular lesions. *J Clin Exp Neuropsychol*. Dec 1990;12(6):857-872.
- 285. Larrabee GJ, Trahan DE, Curtiss G. Construct validity of the Continuous Visual Memory Test. *Arch Clin Neuropsychol.* Oct 1992;7(5):395-405.
- 286. Paolo AM, Troster AI, Ryan JJ. Test-retest stability of the Continuous Visual Memory Test in elderly persons. Arch Clin Neuropsychol. Oct 1998;13(7):617-621.
- 287. Paolo AM, Troster AI, Ryan JJ. Continuous Visual Memory Test performance in healthy persons 60 to 94 years of age. *Arch Clin Neuropsychol.* May 1998;13(4):333-337.
- 288. Snitz BE, Roman DD, Beniak TE. Efficacy of the Continuous Visual Memory Test in lateralizing temporal lobe dysfunction in chronic complex-partial epilepsy. *J Clin Exp Neuropsychol*. Oct 1996;18(5):747-754.
- 289. Hall S, Pinkston SL, Szalda-Petree AC, Coronis AR. The performance of healthy older adults on the Continuous Visual Memory Test and the Visual-Motor Integration Test: preliminary findings. *J Clin Psychol*. Jul 1996;52(4):449-454.
- 290. Harker KT, Connolly JF. Assessment of visual working memory using eventrelated potentials. *Clinical neurophysiology : official journal of the International Federation of Clinical Neurophysiology.* Nov 2007;118(11):2479-2488.
- 291. Banos JH, Dickson AL, Greer T. A computer-assisted administration of the Continuous Visual Memory Test. *Clin Neuropsychol.* Dec 2001;15(4):551-555.
- 292. Retzlaff PD, Morris GL. Event-related potentials during the Continuous Visual Memory Test. *J Clin Psychol.* Jan 1996;52(1):43-47.
- 293. Woods AJ, Hamilton, et al., . Space, time, and causaltiy in the human brain. *Neuroimage*. 2014;in press.
- 294. Woods AJ, Lehet M, Chatterjee A. Context modulates the contribution of time and space in causal inference. *Front Psychol.* 2012;3:371.
- 295. Provencher SW. Automatic quantitation of localized in vivo 1H spectra with LCModel. *NMR in biomedicine*. Jun 2001;14(4):260-264.

- 296. Fischl B, Dale AM. Measuring the thickness of the human cerebral cortex from magnetic resonance images. *Proceedings of the National Academy of Sciences of the United States of America*. Sep 26 2000;97(20):11050-11055.
- 297. Fischl B, Sereno MI, Dale AM. Cortical surface-based analysis. II: Inflation, flattening, and a surface-based coordinate system. *Neuroimage*. Feb 1999;9(2):195-207.
- 298. Fischl B, Sereno MI, Tootell RB, Dale AM. High-resolution intersubject averaging and a coordinate system for the cortical surface. *Human brain mapping*. 1999;8(4):272-284.
- 299. Andrade KC, Pontes-Neto OM, Leite JP, Santos AC, Baffa O, de Araujo DB. Quantitative aspects of brain perfusion dynamic induced by BOLD fMRI. *Arq Neuropsiquiatr.* Dec 2006;64(4):895-898.
- 300. Leoni RF, Mazzeto-Betti KC, Andrade KC, de Araujo DB. Quantitative evaluation of hemodynamic response after hypercapnia among different brain territories by fMRI. *Neuroimage*. Jul 15 2008;41(4):1192-1198.
- 301. Kim SG, Rostrup E, Larsson HB, Ogawa S, Paulson OB. Determination of relative CMRO2 from CBF and BOLD changes: significant increase of oxygen consumption rate during visual stimulation. *Magn Reson Med.* Jun 1999;41(6):1152-1161.
- 302. Kastrup A, Kruger G, Glover GH, Neumann-Haefelin T, Moseley ME. Regional variability of cerebral blood oxygenation response to hypercapnia. *Neuroimage*. Dec 1999;10(6):675-681.
- 303. Posse S, Kemna LJ, Elghahwagi B, Wiese S, Kiselev VG. Effect of graded hypoand hypercapnia on fMRI contrast in visual cortex: quantification of T(\*)(2) changes by multiecho EPI. *Magn Reson Med.* Aug 2001;46(2):264-271.
- 304. Lezak MD. Neuropsychological assessment in behavioral toxicology--developing techniques and interpretative issues. *Scandinavian journal of work, environment & health.* 1984;10 Suppl 1:25-29.
- 305. DiGirolamo GJ, Kramer AF, Barad V, et al. General and task-specific frontal lobe recruitment in older adults during executive processes: a fMRI investigation of task-switching. *Neuroreport*. Jul 3 2001;12(9):2065-2071.
- 306. Gross AL, Rebok GW, Brandt J, Tommet D, Marsiske M, Jones RN. Modeling learning and memory using verbal learning tests: results from ACTIVE. *The journals of gerontology. Series B, Psychological sciences and social sciences.* Mar 2013;68(2):153-167.
- 307. Gunstad J, Cohen RA, Paul RH, Luyster FS, Gordon E. Age effects in time estimation: relationship to frontal brain morphometry. *Journal of integrative neuroscience*. Mar 2006;5(1):75-87.
- 308. Jones RN, Rosenberg AL, Morris JN, et al. A growth curve model of learning acquisition among cognitively normal older adults. *Experimental aging research*. Jul-Sep 2005;31(3):291-312.
- 309. Okonkwo OC, Cohen RA, Gunstad J, Tremont G, Alosco ML, Poppas A. Longitudinal trajectories of cognitive decline among older adults with cardiovascular disease. *Cerebrovasc Dis.* 2010;30(4):362-373.

- 310. Paul RH, Brickman AM, Cohen RA, et al. Cognitive status of young and older cigarette smokers: data from the international brain database. *J Clin Neurosci*. May 2006;13(4):457-465.
- 311. Roller CA, Cohen HS, Kimball KT, Bloomberg JJ. Effects of normal aging on visuo-motor plasticity. *Neurobiol Aging*. Jan-Feb 2002;23(1):117-123.
- 312. Woods AJ, Mark VW, Pitts AC, Mennemeier M. Pervasive cognitive impairment in acute rehabilitation inpatients without brain injury. *PM & R : the journal of injury, function, and rehabilitation.* May 2011;3(5):426-432; quiz 432.
- 313. Zimerman M, Nitsch M, Giraux P, Gerloff C, Cohen LG, Hummel FC. Neuroenhancement of the aging brain: restoring skill acquisition in old subjects. *Ann Neurol.* Jan 2013;73(1):10-15.
- 314. Zlatar ZZ, Towler S, McGregor KM, et al. Functional language networks in sedentary and physically active older adults. *J Int Neuropsychol Soc.* Jul 2013;19(6):625-634.
- 315. Taha J, Czaja SJ, Sharit J, Morrow DG. Factors affecting usage of a personal health record (PHR) to manage health. *Psychology and aging*. Dec 2013;28(4):1124-1139.
- 316. Sharit J, Czaja SJ, Nair S, Lee CC. Effects of age, speech rate, and environmental support in using telephone voice menu systems. *Hum Factors*. Summer 2003;45(2):234-251.
- 317. Baecke JA, Burema J, Frijters JE. A short questionnaire for the measurement of habitual physical activity in epidemiological studies. *Am J Clin Nutr.* Nov 1982;36(5):936-942.
- 318. Richardson MT, Ainsworth BE, Wu HC, Jacobs DR, Jr., Leon AS. Ability of the Atherosclerosis Risk in Communities (ARIC)/Baecke Questionnaire to assess leisure-time physical activity. *International journal of epidemiology.* Aug 1995;24(4):685-693.
- 319. Philippaerts RM, Westerterp KR, Lefevre J. Doubly labelled water validation of three physical activity questionnaires. *International journal of sports medicine*. Jul 1999;20(5):284-289.
- 320. Philippaerts RM, Lefevre J. Reliability and validity of three physical activity questionnaires in Flemish males. *American journal of epidemiology.* May 15 1998;147(10):982-990.
- 321. Cella D, Riley W, Stone A, et al. The Patient-Reported Outcomes Measurement Information System (PROMIS) developed and tested its first wave of adult self-reported health outcome item banks: 2005-2008. *Journal of clinical epidemiology*. Nov 2010;63(11):1179-1194.
- 322. Magasi S, Ryan G, Revicki D, et al. Content validity of patient-reported outcome measures: perspectives from a PROMIS meeting. *Quality of life research: an international journal of quality of life aspects of treatment, care and rehabilitation.* Jun 2012;21(5):739-746.
- 323. Tucker CA, Cieza A, Riley AW, et al. Concept Analysis of the Patient Reported Outcomes Measurement Information System (PROMIS) and the International Classification of Functioning, Disability and Health (ICF). Quality of life research: an international journal of quality of life aspects of treatment, care and rehabilitation. Feb 6 2014.

| 324. | Reeve BB, Hays RD, Bjorner JB, et al. Psychometric evaluation and calibration of health-related quality of life item banks: plans for the Patient-Reported Outcomes Measurement Information System (PROMIS). <i>Medical care</i> . May 2007;45(5 Suppl 1):S22-31. |
|---|---|